

#### **UVA CENTER FOR DIABETES TECHNOLOGY**

# Adapting Diabetes Treatment Expert Systems to Patient's Expectations and Psychobehavioral Characteristics in Type 1 Diabetes

**Protocol Chair** 

Marc Breton, PhD

University of Virginia

Center for Diabetes Technology

Version Number: v2.0

05-Oct-2021



# **KEY ROLES**

| Protocol Principal Investigator | |
|---|---|
| Name, degree | Marc Breton, Ph.D. |
| Institution Name | University of Virginia Center for Diabetes Technology |

DSS-2\_05-Oct-2021 



# **PROTOCOL VERSION HISTORY**

| Version<br>Number | Author(s) | Approver | Effective<br>Date | Revision Description |
|---|---|---|---|---|
| 1.0 | | | 24-Apr-2020 | Original Protocol |
| 1.1 | Mary Oliveri | Mary Oliveri | 20-May-<br>2020 | Added • Demographic Data Survey added at screening |
| 1.2 | Mary Oliveri | | 03-Aug-2020 | <ul> <li>Full Board Revisions:</li> <li>Clarified that participants may contact the study team at any time during the study to report adverse events (Section 5.1.1 5.3.2, 6.4.3, 6.6.3, 7.6.3).</li> <li>Corrected erroneous sentence referencing DHHS 46.405 (section 10.3).</li> <li>Corrected bullet formatting (section 12.3.2).</li> <li>Removed references to Medical Monitor throughout protocol.</li> <li>Added references to Data Safety Monitoring Board (section 12.10).</li> </ul> |
| 1.3 | Jon Olson | Mary Oliveri | 08-Nov-2020 | <ul> <li>Study Team modifications:</li> <li>Physical examination (may use a medical record within the past 6 months)</li> <li>Weight, height (participant may self-report this information)</li> <li>Vital signs including measurement of blood pressure and pulse (may use a medical record within the past 6 months)</li> <li>Participants will have the option to be given a receiver from the study team for medical needs.</li> </ul> |
| 1.4 | Jon Olson | Mary Oliveri | 22-Jan-2021 | <ul> <li>DSMB Request:</li> <li>If applicable, subjects will have a pregnancy test between phases (section 6.4).</li> </ul> |
| 2.0 | Mary Oliveri | Marc Breton, Ralf<br>Nass | 05-Oct-2021 | Study Team Modifications: • Modified HbA1c limit to HbA1c 6.0-11.0%, inclusive (section 3.3)Edited Sensor Augmented Pump Therapy (SAP) to Sensor |

DSS-2\_05-Oct-2021 



| Augmented Mode (SAM) throughout the document Deleted inclusion of carbohydrate counting (section 3.3) Added NPH insulin as study exclusion (section 3.4) Added Post-Screening Assessment section describing participant requirements (section 3.5) Clarified Training visit definition (Chapter 4)Clarified pump and MDI training issues (section 4.1.2, 4.1.3) Study physician may add up to two weeks to CGM run-in period (section 5.2.1) Revised Figure 4 and Figure 5 |
|---|
|---|

DSS-2\_05-Oct-2021 



#### SITE PRINCIPAL INVESTIGATOR STATEMENT OF COMPLIANCE

Protocol Title: Adapting Diabetes Treatment Expert Systems to Patient's Expectations and Psychobehavioral Characteristics in Type 1 Diabetes

Protocol Version/Date: v2.0/05-Oct-2021

I have written the protocol specified above. In my formal capacity as a Site Principal Investigator, my duties include ensuring the safety of the study participants enrolled under my supervision. It is understood that all information pertaining to the study will be held strictly confidential and that this confidentiality requirement applies to all study staff at this site.

This trial will be carried out in accordance with ICH E6 Good Clinical Practice (GCP) and as required by the following: United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812).

As the Principal Investigator, I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), or other approved Ethics Committee, except where necessary to eliminate an immediate hazard(s) to the trial participants.

All key personnel (all individuals responsible for the design and conduct of this trial) have completed Human Participants Protection Training and Good Clinical Practice Training. Further, I agree to ensure that all staff members involved in the conduct of this study are informed about their obligations in meeting the above commitments.

| Investigator's Signature | Date: | / | / |
|-----------------------------------|-------|---|---|
| Investigator's Name: | | | |
| Site Name: University of Virginia | | | |

Dec. 2 of 04 2024



# **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|--------------|-------------------------------------------|
| API | Application Programming Interface |
| ATI | Acceptance and Trust Index |
| BG | Blood Glucose |
| BT/BTLE | Bluetooth, Bluetooth low energy |
| CR | Carbohydrate Ratio |
| CLC | Closed-Loop Control |
| ССБМ | Continuous Glucose Monitor |
| CSII | Continuous Subcutaneous Insulin Injection |
| cv | Coefficient of Variation |
| DiAs | Diabetes Assistant |
| DCCT | Diabetes Control and Complications Trial |
| DKA | Diabetic Ketoacidosis |
| DSS | Decision Support System |
| DWM | DiAs Web Monitoring |
| eA1c | Estimated Hemoglobin A1c |
| EMA | Ecological Momentary Assessment |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GLM | General Linear Models |
| GV | Glucose Variability |
| HbA1c | Hemoglobin A1c |
| HBGI | High Blood Glucose Index |
| НТТР | Hypertext Transfer Protocol |
| IDE | Investigational Device Exemption |
| IOB | Insulin-on-Board |
| ISF | Insulin Sensitivity Factor |
| JSON | JavaScript Object Notation |
| LBGI | Low Blood Glucose Index |
| NIH | National Institutes of Health |
| PF | Personalized Feedback |
| POC | Point-of-Care |

DSS-2\_05-Oct-2021 



| QC | Quality Control |
|----------|----------------------------------|
| QOL | Quality of Life |
| REST-ful | Representational State Transfer |
| SAM | Sensor Augmented Mode |
| SAP | Sensor-Augmented Pump therapy |
| SH | Severe Hypoglycemia |
| SI | Insulin Sensitivity |
| SMBG | Self-Monitoring of Blood Glucose |
| T1DM | Type 1 Diabetes Mellitus |
| T2DM | Type 2 Diabetes Mellitus |
| UI | User Interface |
| URL | Uniform Resource Locator |
| XML | Extensible Markup Language |

DSS-2\_05-Oct-2021 



# **PROTOCOL SUMMARY**

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | Adapting Diabetes Treatment Expert Systems to Patient's Expectations and Psychobehavioral Characteristics in Type 1 Diabetes |
| Investigational Device | CGM-based Personalized Feedback (PF) and Decision Support System (DSS) |
| Objectives | Aim 1 (control of GV) We will confirm and contrast the efficacy of two previously designed technological interventions – Personalized Feedback (PF) and Decision Support System (DSS) - in reducing glucose variability (GV) in Type 1 Diabetes Mellitus (T1DM) during a 6-month randomized crossover clinical trial. |
| | <b>Aim 2</b> (personalization of treatment policy) We hypothesize that the participants in this study will have technology intervention preferences (e.g. PF or DSS) that can be predicted by key psychosocial and behavioral parameters and are prognostic of the level of GV control achievable by the intervention. |
| | <b>Aim 3</b> (monitoring of treatment policy) Finally, we propose to define a novel, measurable, technology Acceptance and Trust Index (ATI), passively observing and recording user-system interactions, and validate this new index using active Ecological Momentary Assessment (EMA) to track user subjective response to DSS. |
| Study Design | This is a randomized crossover study in T1DM adults designed to demonstrate the efficacy of personalized feedback (PF) and decision support (DSS) over sensor-augmented mode (SAM) therapy and to establish relationships between the level of glucose variability (GV) control achievable by the intervention and individual psycho-behavioral characteristics. |
| Number of Sites | 1 |
| Outcomes | A key advantage of the proposed study design (beyond the optimal statistical power) is the possibility to explore the glucose control and psycho-behavioral impact of features being added and/or enhanced with prescriptive components (DSS), vs. features being limited to information (PF) or even removed (SAM). |
| Population | Key Inclusion Criteria Age 18 years and older T1DM diagnosis for at least 1 year Established insulin parameters Key Exclusion Criteria d Hemoglobin A1c 6.0-11.0%, inclusive |
| Sample Size | Enrollment will proceed with the goal of completing 4 cohorts of about 25 participants each (expected retention 20 per cohort) |
| Treatment Groups | <ul> <li>De-escalation (DSS→PF→SAM)</li> <li>Escalation (SAM→PF→DSS)</li> </ul> |
| Participant Duration | The study duration for each participant is approximately 7 months. |
| Protocol Overview/Synopsis | Four cohorts of about 25 participants each (expected retention 20 per cohort). Each cohort will continue for ~7 months. Following recruitment, screening, and a run-in period of SAM, participants will be randomized into one of two groups: escalation vs. de-escalation of devices and function. Each treatment modality (SAM, PF, DSS) will continue for about 8 weeks, with the last 4 weeks used to assess GV from CGM data. |

DSS-2\_05-Oct-2021 

# STUDY VISITS AND PROCEDURES SCHEDULE

| | Visit 1<br>Screening<br>and<br>Questionnaires | Visit 2<br>Study Device<br>and<br>Procedures<br>Training | SAM<br>Run-in | Visit 3 Eligibility Assessment, Randomization and Training | DiAs Use<br>in Phase 1<br>Mode | Visit 4<br>Phase 2<br>Initiation | DiAs Use<br>in Phase 2<br>Mode | Visit 5<br>Phase 3<br>Initiation | DiAs Use<br>in Phase 3<br>Mode | Visit 6<br>Study<br>Exit | Visit 7<br>Post<br>Study<br>Check in |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Location | Clinic | Clinic | Home x<br>2-4<br>weeks | Web<br>Conference<br>or Clinic | Home x<br>8 weeks | Web<br>Conference<br>or Clinic | Home x<br>8 weeks | Web<br>Conference<br>or Clinic | Home x<br>8 weeks | Phone<br>or<br>Clinic | Phone<br>or<br>Clinic |
| Informed Consent | Х | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | |
| Medications | Х | | | | | | | | | | |
| Physical Exam (including vital signs, height/weight) | Х | | | | | | | | | | |
| Pregnancy Test (if childbearing potential) | X | | | | | Х | | Х | | | |
| Blood Testing: TSH, CMP<br>(additional labs as<br>necessary) | х | | | | | | | | | | |
| Questionnaires | Х | | Х | Х | Х | Х | Х | Х | Х | Х | |
| Equipment Training | | Х | | | | | | | | | |
| DiAs in SAM Training | | Х | | | | | | | | | |
| Glycemic Treatment<br>Guidelines Training | | Х | | | | | | | | | |
| Glucagon Emergency Kit<br>Training | | Х | | | | | | | | | |
| Use of DiAs in SAM | | | Х | | | | | | | | |
| Eligibility Assessment | | | | Х | | | | | | | |
| AE Assessment | | | | Х | | Х | | Х | | Χ | |
| Randomization | | | | Х | | | | | | | |
| DiAs Phase 1 Mode Training | | | | Х | | | | | | | |
| EMA Training | | | | Х | | | | | | | |

DSS-2\_05-Oct-2021 

| | Visit 1 Screening and Questionnaires Visit 1 Screening and Questionnaires | Visit 2 Study Device and Procedures Training Visit 2 Study Device and Procedures Training | SAM<br>Run-in<br>SAM<br>Run-in | Visit 3 Eligibility Assessment, Randomization and Training Visit 3 Eligibility Assessment, Randomization and Training | DiAs Use<br>in Phase 1<br>Mode<br>DiAs Use<br>in Phase 1<br>Mode | Visit 4 Phase 2 Initiation Visit 4 Phase 2 Initiation | DiAs Use<br>in Phase 2<br>Mode<br>DiAs Use<br>in Phase 2<br>Mode | Visit 5 Phase 3 Initiation Visit 5 Phase 3 Initiation | DiAs Use<br>in Phase 3<br>Mode<br>DiAs Use<br>in Phase 3<br>Mode | Visit 6<br>Study<br>Exit<br>Visit 6<br>Study<br>Exit | Visit 7 Post Study Check in Visit 7 Post Study Check in |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Location | Clinic | Clinic | Home x<br>2-4<br>weeks | Web<br>Conference<br>or Clinic | Home x 8<br>weeks | Web<br>Conference<br>or Clinic | Home x 8<br>weeks | Web<br>Conference<br>or Clinic | Home x 8<br>weeks | Phone<br>or Clinic | Phone<br>or Clinic |
| Use of DiAs in Phase 1<br>Mode | | | | | Х | | | | | | |
| EMA Surveys | | | | | х | | х | | х | | |
| DiAs Phase 2 Mode Training | | | | | | Х | | | | | |
| Use of DiAs in Phase 2<br>Mode | | | | | | | Х | | | | |
| DiAs Phase 3 Mode Training | | | | | | | | Х | | | |
| Use of DiAs in Phase 3<br>Mode | | | | | | | | | Х | | |
| Review diabetes management & AEs | | | | x | | X | | Х | | Х | Х |

DSS-2\_05-Oct-2021 

# **Table of Contents**

1

| 2 | Chapter | 1 Background | 15 |
|----|---------|-----------------------------------------------|----|
| 3 | 1.1. | Introduction | 15 |
| 4 | 1.2. | Specific Aims | 23 |
| 5 | 1.3. | Outcomes | 24 |
| 6 | 1.4. | Study Design | 27 |
| 7 | 1.5. | Study Participants | 28 |
| 8 | 1.6. | Clinical Sites | 28 |
| 9 | Chapter | · 2 Study Devices | 29 |
| 10 | 2.1. | Diabetes Assistant (DiAs) | 29 |
| 11 | 2.2. | Insulin Pump | 29 |
| 12 | 2.3. | Continuous Glucose Monitor (CGM) | 29 |
| 13 | 2.4. | Ketone Meter and Strips | 29 |
| 14 | Chapter | · 3 Study Screening | 30 |
| 15 | 3.1. | Informed Consent and Authorization Procedures | 30 |
| 16 | 3.2. | Visit 1 - Eligibility Screening Procedures | 30 |
| 17 | 3.3. | Participant Inclusion Criteria | 31 |
| 18 | 3.4. | Participant Exclusion Criteria | 32 |
| 19 | 3.5. | Post-screening assessments | 33 |
| 20 | Chapter | · 4 Training Visit | 34 |
| 21 | 4.1. | Visit 2 - Study Equipment | 34 |
| 22 | 4.2. | Ecological Momentary Assessment Training | 36 |
| 23 | 4.3. | Glucagon Emergency Kit | 36 |
| 24 | Chapter | · 5 Study Procedures | 37 |
| 25 | 5.1. | Study Contacts | 37 |

| 5.2. | Sensor-Augmented Mode (SAM) Run-in Period | 37 |
|--------|--------------------------------------------------------------|----|
| 5.3. | Visit 3 – Eligibility Assessment, Randomization and Training | 38 |
| Chapte | er 6 Study Procedures - Escalation | 39 |
| 6.2. | Sensor Augmented Mode | 39 |
| 6.3. | Home Use of DiAs in Phase 1 Mode | 39 |
| 6.4. | Visit 4 – Phase 2 Initiation | 40 |
| 6.5. | Home Use of DiAs in Phase 2 Mode | 41 |
| 6.6. | Visit 5 – Phase 3 Initiation | 42 |
| 6.7. | Home Use of DiAs in Phase 3 Mode | 43 |
| 6.8. | Visit 6 - Study Exit | 43 |
| 6.9. | Post Study Check-In Visit (Visit 7) | 44 |
| Chapte | er 7 Study Procedures – De-Escalation | 45 |
| 7.1. | Randomization to De-Escalation | 45 |
| 7.2. | Training on Phase 1 DiAs Mode | 45 |
| 7.3. | Home Use of DiAs in Phase 1 Mode | 46 |
| 7.4. | Visit 4 – Phase 2 Initiation | 46 |
| 7.5. | Home Use of DiAs in Phase 2 Mode | 47 |
| 7.6. | Visit 5 – Phase 3 Initiation | 48 |
| 7.7. | Home Use of DiAs in Phase 3 Mode | 48 |
| 7.8. | Visit 6 - Study Exit | 49 |
| 7.9. | Post Study Check-In Visit (Visit 7) | 50 |
| Chapte | er 8 Testing Procedures | 51 |
| 8.1. | Laboratory / Point of Care Testing | 51 |
| Chapte | er 9 Questionnaires & Ecological Momentary Analysis | 52 |
| 9.1. | Diabetes Specific Personality Questionnaire | 52 |
| 9.2. | ABACUS | 52 |

| 2 | 9.3. | Diabetes Locus of Control | 52 |
|---|---|---|---|
| 3 | 9.4. | Confidence in Diabetes Self-Care Scale | 52 |
| 4 | 9.5. | Clarke's Hypoglycemia Awareness Scale | 53 |
| 5 | 9.6. | The Diabetes Distress Scale | 53 |
| ô | 9.7. | Hypoglycemia Fear Survey | 53 |
| 7 | 9.8. | Hyperglycemia Avoidance Scale | 53 |
| 3 | 9.9. | Pittsburgh Sleep Quality Index | 54 |
| 9 | 9.10. | Technology Acceptance and Expectations Survey (burdens subscale only) | 54 |
| ) | 9.11. | INSPIRE (revised for DSS) | 54 |
| L | 9.12. | Ecological Momentary Analysis (EMA) | 54 |
| 2 | 9.13. | Questionnaire Schedule | 56 |
| 3 | Chapter | 10 Risks, Benefits, and Risk Assessment | 57 |
| | 10.1. | Potential Risks and Benefits of the Investigational Device | 57 |
| | 10.2. | Potential Benefits | 59 |
| | 10.3. | Risk Assessment | 59 |
| | 10.4. | General Considerations | 59 |
| | Chapter | 11 Device Cleaning Instructions | 61 |
| ı | Chapter | 12 Adverse Events, Device Issues, and Stopping Rules | 62 |
| ) | 12.1. | Definitions | 62 |
| L | 12.2. | Protocol Deviations | 63 |
| <u>)</u> | 12.3. | Reportable Events | 63 |
| } | 12.4. | Relationship of Adverse Event to Study Device | 64 |
| ļ | 12.5. | Intensity of Adverse Event | 65 |
| , | 12.6. | Coding of Adverse Events | 65 |
| | 12.7. | Outcome of Adverse Events | 65 |
| , | 12.8. | Reportable Device Issues | 66 |

| 78 | 12.9. | Timing of Event Reporting | 67 |
|---|---|---|---|
| 79 | 12.10. | Data and Safety Monitoring Board | 67 |
| 80 | 12.11. | Stopping Criteria | 68 |
| 81 | 12.12. | Independent Safety Oversight | 68 |
| 82 | Chapter 1 | .3 Miscellaneous Considerations | 69 |
| 83 | 13.1. | Prohibited Medications, Treatments, and Procedures | 69 |
| 84 | 13.2. | Participant Withdrawal | 69 |
| 85 | 13.3. | Confidentiality | 69 |
| 86 | Chapter 1 | .4 Statistical Consideration | 70 |
| 87 | 14.1. | Design and Randomization | 70 |
| 88 | 14.2. | Sample Size | 70 |
| 89 | 14.3. | Outcome Measures | 71 |
| 90 | 14.4. | Exploration of the effect of treatment escalation vs. de-escalation | 72 |
| 91 | 14.5. | Psychological and Behavioral Questionnaires | 72 |
| 92 | 14.6. | Baseline Descriptive Statistics | 72 |
| 93 | 14.7. | Device Issues | 72 |
| 94 | Chapter 1 | .5 Data Collection and Monitoring | 73 |
| 95 | 15.1. | Case Report Forms and Device Data | 73 |
| 96 | 15.2. | Study Records Retention | 73 |
| 97 | Chapter 1 | .6 Ethics/Protection of Human Participants | 74 |
| 98 | 16.1. | Ethics Standard | 74 |
| 99 | 16.2. | Institutional Review Boards | 74 |
| 100 | 16.3. | Informed Consent Procedures and Documentation | 74 |
| 101 | 16.4. | Participant and Data Confidentiality | 74 |
| 102 | Chapter 1 | .7 References | 76 |

103

104

105

106

115

116

117118

119

120

121

122

123

124

125

126

127

128

129

130

131

132133

# Chapter 1 Background

#### 1.1. Introduction

#### 107 **1.1.1.** Significance

Type 1 diabetes mellitus (T1DM) is an autoimmune condition resulting in absolute insulin deficiency and a life-long need for insulin replacement [1]. Glycemic control in T1DM remains a challenge, despite the availability of modern insulin analogs [2], the improving accuracy of glucose monitoring [3-4], and the widening use of intensive insulin therapy. While new technologies have proven benefits in avoiding diabetes related complications [5] and may have reduced excess mortality in some populations [6], excess mortality and complication rates remain significantly higher in T1DM when compared to the general population [7-8].

Glucose variability (GV) in T1DM is typically at the root of clinicians' inability to safely achieve near-normal average glycemia, as reflected by hemoglobin A1c (HbA1c) [9]. While target HbA1c values of 7% or less result in decreased risk of micro- and macrovascular complications [10-13], the risk for severe hypoglycemia (SH) increases with tightening glycemic control [14-16]. Consequently, hypoglycemia has been implicated as the primary barrier to optimal control [17-18]. Thus, individuals with T1DM face a life-long optimization challenge: reduce average glucose levels and postprandial hyperglycemia while simultaneously avoiding hypoglycemia. A strategy for achieving such an optimization can only be effective if it reduces GV. This is because bringing average glycemia down is only possible if GV is constrained – otherwise blood glucose (BG) fluctuations would inevitably enter the range of hypoglycemia. However, averages and HbA1c fail to capture GV and the attendant risks associated with extremes of hypo- and hyperglycemia. Indeed, in addition to establishing HbA1c as the gold standard for average glycemic control, the Diabetes Control and Complications Trial (DCCT) concluded that: "HbA1c is not the most complete expression of the degree of glycemia. Other features of diabetic glucose control, which are not reflected by HbA1c, may add to, or modify the risk of complications. For example, "the risk of complications may be highly dependent on the extent of postprandial glycemic excursions" [19]. Thus, more recent studies increasingly focused on the variability of BG fluctuations as an independent risk factor for diabetes complications [9, 20-21], particularly cardiovascular disease [22-25].

DSS-2\_05-Oct-2021 

134

135

136

137138

139

140

141

142

143

144

145

146147

148

149150

151152

153

154

155

156157

158

159

160

161

162

163164

165

166

167168

Intensive insulin therapy: Introduced in the 1980s, intensive insulin treatment by multiple daily injections (MDI) or use of continuous subcutaneous insulin infusion (CSII), typically includes basal insulin administered to cover the overnight and fasting periods and bolus insulin given with meals to cover carbohydrate consumption and to correct postprandial hyperglycemia, in an attempt to mimic insulin secretion in health [26]. Advanced insulin therapy relies on key individual parameters such as basal rate, carbohydrate ratio (CR) and insulin sensitivity factor (ISF) [26]. Evidence-based resources are available to patients to control their insulin intake and schedules, and clinicians to initiate and maintain CSII therapy by selecting appropriate basal rates, carbohydrate ratios, and insulin sensitivity factor patterns [27].

Expert systems and Control of Glucose Variability: Periodic adjustments of basal rate, CR, and ISF patterns are needed based on review of self-monitoring blood glucose (SMBG) profiles, or continuous glucose monitoring (CGM). If a pattern is identified, optimized insulin dosing parameters are calculated and implemented. This can be a time-consuming and onerous task, requiring data to be downloaded from multiple devices and often subjectively evaluated. Information technology is increasingly playing a positive role in improving the management of chronic conditions [28-29], including diabetes [30]. For example, in T1DM, telemedicine and online patient support has shown promising results [31-32]; and retrospectively linking behavior to glycemic outcomes has proven effective as well [33]. With improvements in SMBG and CGM technologies, a growing appreciation of the quantitative (algorithmic) aspect of the management of T1DM has led to new tools for remote patient monitoring, data aggregation and visualization [34]. Early research has developed algorithms for titrating individual insulin treatment parameters, including iterative learning approaches such as 'run-to-run' with structured SMBG [35-39]. Insulin titration and dosing tools for type 2 diabetes are beginning to enter the marketplace [40], mostly using SMBG. Today, researchers are actively working on CGM-based decision support for T1DM [26, 41-44], capable of providing specific feedback to the clinician regarding suggested therapy changes. These expert systems have the potential to streamline clinic visits and facilitate collaborative patient-centered interactions, but in their most advanced form, they deliver advice directly to the patient [41], reducing burden and uncertainty when making self-management decisions.

<u>Automated Insulin Delivery:</u> Closed loop control (CLC) technology (i.e. artificial pancreas or AP), involves the pairing of CGM with CSII (insulin pump) via a closed loop control algorithm which automatically adjusts insulin infusion in real-time [45]. In the past decade, AP studies have advanced from short-term inpatient studies [46], to long-term clinical trials in free-living conditions using wearable wireless automated AP systems [47]. Our AP studies have enrolled >450 T1DM patients, who used our smartphone-based system for over 280,000 hours.

DSS-2\_05-Oct-2021 

169 Algorithmic advances and computational platforms from these efforts are at the core of this

170 investigation.

179

180

183

184

187

193

171 Smartphone based data acquisition and advice delivery platforms: This investigation brings

172 together two key pieces of mobile technology to advance T1DM treatment: The Diabetes

173 Assistant (DiAs) and Ecological Momentary Assessment (EMA).

<u>Diabetes Assistant (DiAs):</u> The Diabetes Assistant (DiAs) 174 175 [48-49] platform is a smartphone-based, modular,

portable device developed at the University of Virginia

176 (UVa), in collaboration with the University of Montpellier

177

178 (Figure 1). DiAs operates on a commercial phone, using a

specifically modified Android operating system, to enable wireless communication with satellite devices like insulin

pumps, CGMs, and any medical device using a standard

181 wireless protocol like BT or BTLE. Its modular architecture 182

allows different control modules to be swapped in real

time, enabling either automated control (CLC) or expert-

185 decision support systems. The DiAs platform also

186 integrates automated data transfer to a secured server,

enabling cloud functionalities such as remote monitoring

188 and patient specific adaptation of treatment [50]. DiAs is

189 filed with the FDA (MAF 2109) and has been approved for

190 use by adults, adolescents, and children with T1DM in



192 insulin and cloud applications; it is the most advanced research glucose control platform to date

and has been deployed for months in home CLC trials. DiAs enables the seamless integration and

194 sequential development of modular decision support systems in a form factor assessed by focus

195 groups to be acceptable by people with T1DM.

196 Leveraging EMA to assess user's subjective reactions to the decision support system will enable

197 the first study with such detailed and dynamic investigation of daily trust levels, psychological,

198 and behavioral responses.

199 Remote computation and cloud analytics: DiAs is capable of real-time data transmission to secure

200 remote servers: the DiAs Web Monitoring (DWM) is a suite of functionalities located on a secure

201 server within the UVA Health System network. At its core is a database that receives real-time

202 data about the DiAs status, such as CGM, insulin delivered, connectivity status, and algorithm

203 status. The system is equipped with a dedicated interface to allow for third party applications to



Figure 1: The DiAs system, a mobile Glucose control platform

DSS-2\_05-Oct-2021 

access data stored on the DWM server. It relies on the HTTP protocol and a Representational State Transfer (REST-ful) architecture to provide authenticated users with access to the content of the database, formatted as JSON or XML. The API uses a URL-based system of requests to target and filter the data sent to the client. Several systems are already connected to DWM [50-52].

Impact of technology trust and acceptance in glycemic control: Trust must be earned; it cannot be assumed. The concept of trust plays an important role in an individual's willingness to engage in the use of a medical device. In its basic definition 'trust is to depend or rely on another' [53]. The "other" can be another person or a device. Trust and acceptance incorporate several key constructs i.e. confidence versus fear, satisfaction versus burden, distress versus improved quality of life. Additional factors include perceived usefulness, cost-benefit balance, perceived ease of use, or impact on others as well as oneself (positive and negative) [54-55].

Human factors research indicates that such psychosocial variables play an important role when it comes to technology uptake. In CGM, factors predictive of uptake and effectiveness, include perceived system reliability and ease-of-use [53,56]. Prior CLC research has also shown that clinical trials participants were quick to trust a novel device (CGM, CSII and algorithm), sacrificing personal control over diabetes management to the system, whilst a negative experience impeded trust, contributing to discontinued use. Other studies of CLC systems have found that, when users lack trust, they tend to override the devices, while users who report trust in the system experience decreases in diabetes burden and stress [57]. In general, trust is associated with positive glycemic outcomes and improved psychosocial functioning and quality of life (QOL) [58]. Barriers to trust and continued acceptance include frustration felt when expectations of the system are not met; feelings of being overwhelmed by the amount of information provided, or negative reactions from the social environment e.g. diabetes-related stigma, possibly resulting in a perceived need to explain/justify why a technical device is worn constantly on the body [53]. In addition to patients' perceptions rooted in their previous experience, unrealistic expectations may lead to disappointment and discontinuation of the device.

General 'tech savviness' can also play a role in acceptance in that those more familiar and comfortable with technology may be more willing to trust the system. Furthermore, the time and effort required to invest in building device-related skills, trust and acceptance may be underestimated (and often is), as these range from technical handling to integrating the system information into one's diabetes self-management and everyday living without intrusive disruptions. Therefore, psychological and behavioral factors play a critical role in the acceptance of diabetes technologies and the trust patients put in them. It is crucial to determine the psychosocial and behavioral predictors to uptake and continued use of technology in order to aid

DSS-2\_05-Oct-2021 

identification of those individuals most likely to realize benefits of any intervention as well as those individuals who may require more support to succeed with technology. Additional individual patient's characteristics (e.g. diabetes belief systems and self-management skills) may be predictive of technology acceptance, trust, use, and benefit. At present, little is known about psychological, behavioral and social factors that contribute to diabetes technology adoption and successful use.

- This investigation will determine psychosocial and behavioral predictors of intervention efficacy, providing data and psychological techniques to support future onboarding and successful use of the DSS, as well as validate novel mechanisms to track trust and acceptance, allowing future systems to adapt to the user's needs, minimizing potential burden and lifestyle interference, and ensuing individualized, person-centered support for optimal glycemic and psychosocial/quality of life outcomes.
- **Hypothesis:** We hypothesize that psycho-behavioral factors are likely to influence system acceptance and trust, and ultimately the patients' success in leveraging the device to achieve their individual goals, e.g. better glycemic control with similar burden, or lower treatment burden with similar glycemic control. To our knowledge, no technological intervention has been assessed in terms of which mode of advice or information delivery is most appropriate to a patient's unique characteristics. Thus, the proposed study is the first to map key psycho-behavioral factors to the expert system characteristics that are most beneficial for treatment success.
  - Tracking and Quantifying User/System Interactions: This study merges the expert platform (DiAs) with software designed to detect, record, and contextualize the interactions between the patient and a medical device. This unique combination of established mobile diabetes technology and cutting-edge software previously unrelated to diabetes, will allow: (i) systematically record treatment behaviors; (ii) track user/system interactions, and (iii) accurately quantify the resulting glucose control. The new DiAs-EMA system is a key innovation and a new tool enabling us to study the interplay of technology, behavior, and treatment of diabetes.
- Using a tracking system, the investigators will be able to observe each user of the system; this in turn allows for an internal quantification of the user level of trust and acceptance and its time course.
  - Modular Design of Decision Support Systems: The AP and diabetes expert systems are assembled from independent (but compatible) modules, each performing a specific control or diagnostic function, e.g. prevention of hypoglycemia or postprandial insulin corrections [59-60]. This architecture allowed for sequential testing and clinical deployment of AP and DSS components and provided a structured framework for networks of control systems [60]. This

DSS-2\_05-Oct-2021 

architecture is fundamental to the goals of this project: we plan to further refine and evaluate a layered glucose variability control system activating different modules depending on the stage of the proposed study (PF vs DSS). Moreover, a modular system is inherently capable of graceful degradation-the capacity to ensure safety even if a module fails. Eventually, this architecture would allow the system to adapt its function to maximize system use and adherence, sequentially enabling more advanced functions as patients build trust and integrate DSS in their treatment. The modules to be included in the PF and DSS have been validated in human clinical trials (see 1.1.2 Preliminary Data). These modules include:

- CGM value, trace, and threshold alarms (applicable to SAM & PF & DSS): Similar to commercial real-time CGM (e.g. Dexcom G6), this module informs the user of the current glucose level and how it has changed recently, enabling treatment decisions. Alerts are set by the user to trigger if BG leaves a preset range.
- Hypoglycemia Risk Indicator (PF & DSS): Based on our group's work in the 1990s and the definition of the glycemic risk ranges [61], we have developed short (1-3 hours), medium (1-3 days), and long (1-3 weeks) term hypoglycemia risk indices. Prototypes of these modules have been evaluated clinically (see Preliminary Data).
- Insulin Sensitivity Profile & Indicator (PF & DSS): We have designed an algorithm capable of tracking changes in insulin sensitivity (SI) and creating daily and monthly SI profiles [62]. We additionally validated a real-time SI indicator to inform insulin dosing (e.g. is the patient more or less sensitive than usual?) [41].
- Insulin on Board (PF & DSS): IOB is a key index to avoid insulin stacking and is available to DiAs through its insulin pump connectivity. DiAs uses a common 4-6 hours action curve derived from encoparesis study [63].
- Exercise Advice (DSS): From our modeling work [64], we have derived an advisory module that ensures safety of mild to moderate exercise by predicting whether an exercise bout is likely to result in hypoglycemia and providing a graded carbohydrate supplementation strategy. See clinical validation in [64].
- **Bedtime Advice (DSS):** Similar to the Exercise advisor, this module uses logistic regression and recent data (CGM, insulin and meals) to gauge overnight hypoglycemia risk and provide bedtime carbohydrate advice.
- Smart Bolus Calculator (DSS): DSS supports advanced bolus calculation capable of accounting for several GV factors such as metabolic characteristics (correction based on 45 min predicted glucose to account for insulin delays) and SI fluctuations (insulin sensitivity tracker).
- Automated Treatment Parameter Optimization (DSS): Based on replay simulation technology [42], this optimization routine analyzes the previous 30 days of CGM, insulin, and meal data to provide updated insulin treatment parameters (CR, ISF).

DSS-2\_05-Oct-2021 

#### 1.1.2. Preliminary Data

309

310

311

312

313

314

315

316

317

318

319

320

321

322

323

324

325

326

327

328

329330

331

332333

334

335

336

337

338339

340

341

342343

**SMBG** Information-Based Decision Support (PF, 2006-11): We have shown that automated behavioral feedback delivered in the field by a portable device can optimize glycemic control by reducing HbA1c and/or occurrence of severe hypoglycemia [33]. We tested the effect of an automated system providing real-time estimates of HbA1c, glucose and variability, risk hypoglycemia. For 10 months, 120 adults with T1DM, performed SMBG and received feedback at three increasingly



Figure 2: Results from 1-year automated decision-support intervention based on SMBG data, with 3 levels of feedback to the patient

complex levels (3 months, each): (i) routine SMBG; (ii) estimated HbA1c, hypo risk, and glucose variability; (iii) estimates of symptoms potentially related to hypoglycemia. HbA1c, and hypoglycemia were evaluated at baseline and at the end of each level. This information-based decision-support reduced HbA1c from 8.0 to 7.6%, p=0.001 (effect confined to subjects with baseline HbA1c above 8.0. Incidence of symptomatic moderate/ severe hypoglycemia was reduced from 5.72 to 3.74 episodes/person per month (p=0.019), more prominently for subjects with history of SH or hypoglycemia unaware (*Figure 2*). We therefore concluded that feedback of SMBG data and summary SMBG-based measures can result in improvement in average glycemic control and reduction in moderate/severe hypoglycemia [33]. The system used in this study was an early prototype of the PF developed here but leveraging only SMBG data [33]. This technological limitation necessitated manual input of high measurement frequencies (4-10 SMBG per day). This investigation leverages automatically collected high frequency CGM data to further improve the usability of the PF system, as well as comparing the effect and acceptability of DSS to more prescriptive features.

**Pilot study of Decision Support (DSS, 2012-2017):** The feasibility and safety of a prototype DSS was tested in 15 women and 9 men with T1DM on insulin pump (N=16) or MDI (N=8),

DSS-2\_05-Oct-2021 

NCT02558491. Age was 37±11 years old, average T1DM duration was 21±11 years. Participants were well controlled on average (HbA1c of 7.2±1%). Participants followed a non-blinded randomized crossover design, with two 48-hours observation periods where patients were exposed to a variety of meals and physical activities to challenge their own control strategies and the DSS. DSS was shown to be feasible and safe (no adverse events). Furthermore, GV was significantly improved (primary outcome, CGM coefficient of variation) from 0.36±0.08 during standard of care to 0.33±0.06 using DSS, p=0.045, with maximum effect during daytime. Further GV analysis using the Low and High blood glucose indices (LBGI, HBGI, [65]), confirmed that most of the observed improvement was due to the hypoglycemia-related GV measured by the LBGI: 2.5±2.1 to 1.6±1.3, p=0.042. As depicted in (Figure 3), protection from hypoglycemia was improved significantly while using the DSS: median percent time spent below 70mg/dL was reduced 3.5-fold, from 3.2% to 0.9%, p=0.018, while maintaining average glycemia 155±27mg/dL vs. 155±23mg/dL, p=0.86. [41]



Figure 3: Impact of DSS on exposure to hypoglycemia and average glucose. Control (grey dots and envelop) and Treatment (black dot and dark grey envelop) are linked by the dotted line for each subject.

Ecological Momentary Analysis (EMA): Our research group has a long and prolific history in the use of EMA to study associations between glycemic parameters and psychosocial and behavioral variables. Our original EMA studies were conducted in the 1980s using pen and paper questionnaires completed just before SMBG, 3-5/day over several weeks. We investigated numerous aspects of living with T1D, including idiosyncratic symptoms associated with BG fluctuations [66-67], patient ability to recognize hypo- and hyperglycemia [68-69], adherence to SMBG recommendations, and relationships between BG extremes and mood state [70-71]. In the 1990s handheld personal computer technology replaced paper for the collection and storage of more complex daily diary data with date & time stamps. This technological advance allowed us to investigate relationships between diabetes self-management behaviors and BG patterns, as well as treatment decision-making (e.g. to drive or not when BG is low) [72-75].

DSS-2\_05-Oct-2021 

As technology continued to advance, we were able to program daily diaries to include, not only questionnaires, but also brief cognitive tasks, which could be timed and scored. In a series of studies in the early 2000s [76-79], our group utilized PDAs to investigate cognitive performance in real-world settings at different BG levels in adults with T1DM and T2DM [77] and school-aged children [79]. Additionally, we conducted studies exploring the relationships between glycemic fluctuations and symptoms/moods in patients with T2DM [76] and the ability of young children and their parents to recognize hypoglycemia [78]. Leading to our first DSS system.

Over the past few years, our group has combined EMA approaches with CGM data collection in innovative ways to address clinically important questions regarding relationships between BG levels and behavioral variables, such as the association between psychological stress and BG patterns using CLC algorithms [80]; where we found a small but significant association between stress and glycemic instability. In 2017, we used the EMA approach in a study of the accuracy of Diabetes Alert Dogs, comparing daily diaries of dog alerts to blinded CGM data [81-82]. That study documented that accuracy at detecting hypoglycemia was highly variable across individual dogs and highlighted the need for standardized training and performance. Most recently, our team has completed a clinical trial using EMAs in a sample of older adults (age > 65) and children with T1DM to assess the cognitive impact of CLC; the data collection process was a success, but the analysis is still undergoing, and we expect to publish these results by the end of 2020. In addition to the above studies, our group also has a long history of using EMA approaches to collect preand post-intervention data in clinical trials of behavioral interventions [66-69], as proposed here. Taken together, there is ample evidence of our group's experience and expertise with research using EMA methods.

Based on these pilot results, we propose to move forward with demonstrating the superior efficacy of a CGM-based advisory system in T1DM, as compared to SAM, and with characterizing the impact of psycho-behavioral factors on system performance, which will enable system individualization and lead to automated adaptation of advice delivery to optimize glycemic control and reduce the system's psychological impact.

#### 1.2. Specific Aims

Aim 1 (Control of Glucose Variability) We will confirm and contrast the efficacy of two previously designed technological interventions – Personalized Feedback (PF) and Decision Support System (DSS) - in reducing GV in T1DM during a 6-month randomized crossover clinical trial. This will allow us to show:

DSS-2\_05-Oct-2021 

- 409 Aim 1.1 the superiority of the PF over Sensor-augmented mode (SAM) in controlling GV. PF is a
- 410 system designed to provide patients with actionable information about glucose control in general
- and GV in particular (e.g. estimated HbA1c (eA1c), risk of hypoglycemia, and activity level);
- 412 **Aim 1.2** the superiority of the DSS over SAM in controlling GV. DSS is a CGM-based system that
- 413 includes PF and further assists with treatment recommendations for common metabolic
- 414 challenges;
- 415 Aim 1.3 the overall non-inferiority of DSS over PF intervention to control GV and superiority of
- 416 DSS to maintain tight glycemic control over time (lower variations of GV in time).
- 417 Aim 2 (personalization of treatment policy) We hypothesize that the participants in this study
- 418 will have technology intervention preferences (e.g. PF or DSS) that can be predicted by key
- 419 psychosocial and behavioral parameters and are prognostic of the level of GV control achievable
- 420 by the intervention. We will:
- 421 Aim 2.1 confirm that technology acceptance and trust are predictive of the level of GV control
- 422 achieved during the study (see Aim 1), regardless of the type of DSS system in use. We
- 423 hypothesize that technology acceptance will correlate negatively with GV: i.e. higher technology
- 424 acceptance leads to lower GV;
- 425 **Aim 2.2** explore the impact of technology expectations and experience on the performance of
- 426 each type of technology intervention (SAM, PF, DSS). For example, higher expectation will
- 427 negatively correlate with GV for the SAM treatment, but not the DSS treatment.
- 428 Aim 2.3 assess the correlation between relevant psycho-behavioral traits with the performance
- 429 of PF vs DSS, identifying potential pathways to the corresponding optimal technology-based
- 430 treatment policies.
- 431 **1.3. Outcomes**
- 432 **1.3.1.** Glycemic outcomes
- The primary outcome of this study will be Glucose Variability (GV) as measured by CGM-based
- 434 Coefficient of Variation (CV), as recommended by the International Consensus on Use of
- 435 Continuous Glucose Monitoring. To further characterize glucose control, we will compute other
- 436 CGM Consensus outcomes as well:
- 437 Average
- 438 Percent in different ranges:
- 439 <50 mg/dL
- 440 <54 mg/dL

DSS-2\_05-Oct-2021 

| 441 | 0 | <60 mg/dL |
|-----|---|----------------|
| 442 | 0 | <70 mg/dL |
| 443 | 0 | ≤70-≤180 mg/dL |
| 444 | 0 | >180 mg/dL |
| 445 | 0 | >250 mg/dL |
| 446 | 0 | >300 mg/dL |

 Each modality of treatment will be assessed using the last 4 weeks of CGM recordings, as we expect most of the GV benefits of each intervention to be realized within the first 4 weeks of the intervention, and a minimum of 24 days of data is considered optimal for CGM—based CV determination.

#### 1.3.2. Glucose Variability Reduction Achieved with CGM-based expert systems

General linear models (GLM) (repeated measures ANOVA) will be used to assess the significance of the differences in average response between SAM, PF, and DSS across appropriate CGM-based metrics. The particular design of the clinical study allow for Aims 1.1, 1.2, and 1.3 to each be addressed independently in a randomized crossover analysis, as shown in Figure 4. While the randomized order of the interventions (escalation vs de-escalation) allows for an objective assessment of the average efficacy of each of them, we will introduce the order as a fixed factor to verify if significant study effects can be detected. Finally, we will study the evolution of GV within each modality period: GV and other CGM-based outcomes will be computed bi-weekly (the minimum length of time for precise GV assessment) and entered in a repeated measures GLM analysis; within-subject contrast (linear and polynomial) using 5 repeated measures per condition to explore the evolution of the glycemic outcomes in time; Aim 1.3.



Figure 4: Multiple analyses enabled by study design to address Aim 1.1, 1.2 and 1.3

DSS-2\_05-Oct-2021

#### 1.3.3. Exploration of the effect of treatment escalation vs. de-escalation

A key advantage of the proposed study design (beyond the optimal statistical power) is the possibility to explore the glucose control and psycho-behavioral impact of features being added and/or enhanced with prescriptive components (DSS), vs. features being limited to information (PF) or even removed (SAM). We will perform this analysis by looking at the between factors in the repeated ANOVA analysis, contrasting the escalation group vs. de-escalation group. While not powered, this analysis will provide key insights in the future feature adaptation schemes based on the ATI.

#### 1.3.4. Psychological and Behavioral Questionnaires

As part of Aim 2, we will conduct robust psychosocial analyses of factors important to participant experience. This will examine relevant core constructs of trust, acceptance, satisfaction, confidence as well as fear, worries, distress and burden. Validated and reliable measures will be used to explore psycho-behavioral characteristics and outcomes in addition to specifically adapted measures for SAM and DSS technologies to capture holistic, disease-specific and technology-specific data. These questionnaires will evaluate how specific constructs are predictive of successful glycemic outcomes associated with DSS. These questionnaires will enable us to assess important non-glycemic treatment outcomes that are meaningful to patients including those affecting Quality of Life (QOL) (e.g. fear of hypoglycemia and diabetes distress). To those ends, participants will complete a battery of questionnaires related to diabetes management, treatment satisfaction and QOL at baseline (before system use) and after each treatment modality.

#### 1.3.5. Ecological Momentary Assessment Data Collection

Participants will be trained on the EMA surveys and requirements. During each treatment condition, over the course of 2-3 days every two weeks, the participant will be asked to complete a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per participant during each Phase. The DiAs phone will display a text message containing a link to the survey. Surveys will be triggered at fixed times, including a morning survey ~1h after waking up and an end-of-the-day survey around 8-9 PM. Participants will be able to delay (up to 30 min) or skip (up to 2 per day excluding at wake up) surveys for their convenience. Participants will respond to questions on a 5-point Likert scale (0=Not at All, 4=Extremely). The first Diary for each day will contain two additional items for rating sleep quantity/quality. The Daily Diary questions are intended to assess agreement, trust, treatment satisfaction, diabetes burden, self-efficacy, mood valence, energy level, physical well-being, and concerns about hypo- and hyperglycemia. The first Diary for each day will contain two additional items for rating sleep quantity/quality.

DSS-2\_05-Oct-2021 

#### 1.3.6. Mapping of Psycho-behavioral Characteristics to DSS Preferences and Performance

Baseline assessments of psycho-behavioral traits will be introduced as covariates in the general linear model when analyzing the glycemic performance of each treatment modality (SAM, PF, DSS). Contrasts will be used to study each pair, specifically SAM vs any advisory system. For constructs that can be changed by the intervention itself (e.g. Fear of hypoglycemia) and that are therefore measured after each intervention, we will use repeated measures model with within-subject covariates (MIXED models) to understand their impact on DSS efficacy. This analysis will shed light on the relationship between the efficacy of treatment modality and individual patient characteristics; Aims 2.1 and 2.2

Using the cloud data system, we will isolate patient-system interactions for each advisory module (e.g. eA1c, predictive hypoglycemia alert), and compute for each subject the probability of the interaction to lead to the expected action, and positive glycemic outcomes. These probabilities will then be used as outcome variables in separate analysis to assess whether psycho-behavioral traits are associated with the acceptance of specific advisory functionalities (e.g. Fear of Hypoglycemia could be lowered by the hypoglycemia prediction module); answering **Aim 2.3.** 

#### 1.3.7. Identification and Validation of the Acceptance & Trust Index

Finally, we will use the validated trust and acceptance measures obtained throughout the protocol to validate the dynamic tracking of ATI. The 80 studied subjects will be divided in 4 cohorts of 20, the first 3 groups used to iteratively refine our estimation procedure (interaction quantification and dynamical model parameters) to accurately reproduce acceptance and trust fluctuations. The last group will be used to prospectively demonstrate the correlation between ATI, trust, and acceptance, thereby addressing **Aim 3.2**; retrospectively we will use the finalized method on all 80 participants to compute the auto-correlation between trust and acceptance and ATI and study the ability of ATI to track changes in time; **Aim 3.3**. Such an index, shown to follow the evolution of robustly assessed trust and acceptance (via standard methods) will enable future systems to characterize its interactions with its user, detecting early drop in adherence and disconnect with patient's expectation (fault detection), and potentially associating them with specific functionalities (fault classification), leading to self-adaptations capable of optimizing system use and trust.

#### 1.4. Study Design

This is a randomized crossover study in T1DM designed to demonstrate the efficacy of personalized feedback (PF) and decision support (DSS) over sensor-augmented mode (SAM) therapy and to establish relationships between the level of glucose variability (GV) control achievable by the intervention and individual psycho-behavioral characteristics.

DSS-2\_05-Oct-2021 

We plan to split the study into 4 cohorts of about 25 participants each (expected retention 20 per cohort). Each cohort will continue for ~7 months and will have the structure presented in Figure 5. Following recruitment, screening, and a run-in period of SAM, participants will be randomized into one of two groups: escalation vs. de-escalation of devices and function. Each treatment modality (SAM, PF, DSS) will continue for about 8 weeks, with the last 4 weeks used to assess GV from CGM data.

De-escalation: DSS → PF → SAM Escalation: SAM → PF → DSS



Figure 5: Study design and timeline

#### 1.5. Study Participants

We anticipate recruiting a total of 100 adults aged 18 years and older. An equal numbers of males and females will attempt to be recruited and all racial/ethnic groups will be eligible for participation. Based on our experience in previous studies of this magnitude, we expect that 80% of recruited subjects will complete the entire trial. Enrollment in the study will proceed with the goal of completing approximately 80 subjects. Up to 150 participants may sign the consent form. Eligibility criteria ensure that the subject will be able to fully deploy the technology in this study. Exclusions include any known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.

#### 1.6. Clinical Sites

The study will be performed at the University of Virginia.

DSS-2\_05-Oct-2021 

# **Chapter 2** Study Devices

#### 554 2.1. Diabetes Assistant (DiAs)

- The Diabetes Assistant (DiAs) system which is a medical platform that uses a smart-phone to
- connect to a continuous glucose sensor to insulin pump and run closed-loop control.

#### 557 **2.2.** Insulin Pump

- For CSII participants, the study system will include a modified Tandem t:slim X2 insulin pump
- 559 (Tandem Diabetes Care, Inc., San Diego, CA), capable of communicating wirelessly with DiAs
- 560 (t:AP).

553

#### 561 2.3. Continuous Glucose Monitor (CGM)

- The study CGM will include Dexcom G6® transmitter and sensors (Dexcom, Inc., San Diego, CA)
- 563 connected to the Diabetes Assistant (DiAs).

#### 564 2.4. Ketone Meter and Strips

- 565 Blood ketone levels will be measured using Precision Xtra® meters and strips (Abbott
- 566 Laboratories Inc., Alemeda, CA) in accordance with the manufacturer's labeling. The blood
- 567 glucose meter component of the Precision Xtra® will not be used.

568



569 570

Figure 6: Study Equipment

DSS-2\_05-Oct-2021 

# **Chapter 3** Study Screening

- 572 3.1. Informed Consent and Authorization Procedures
- 573 Before consent has been obtained, participants will be asked inclusion/exclusion criteria
- 574 questions during prescreening to determine study eligibility. Before completing any procedures
- or collecting any data that are not part of usual care, written informed consent will be obtained.
- 576 Potential eligibility may be assessed as part of a routine-care examination.
- A participant is considered enrolled when the informed consent form has been signed by the
- 578 participant and the study team.
- 579 Consenting procedures and documentation is defined in section 16.3.
- Virtual study visits may take the place of all in-person study visits as deemed feasible by the study
- 581 team.

571

- 582 **3.2. Visit 1 Eligibility Screening Procedures**
- After informed consent has been signed, a potential participant will be evaluated for study
- eligibility through the elicitation of a medical history, performance of a physical examination
- by licensed study personnel, blood draw and urine pregnancy testing (if applicable) to screen for
- 586 exclusionary medical conditions.
- 587 The following procedures will be performed/data collected/eligibility criteria checked and
- 588 documented:
- Inclusion and exclusion criteria assessed
- Demographics (address, date of birth, gender, race, ethnicity)
- Contact information
- 592 Diabetic history
- Medical history
- 594 Medications
- Physical examination (may use a medical record within the past 6 months)
- Weight, height (participant may self-report this information)
- Vital signs including measurement of blood pressure and pulse (may use a medical record within the past 6 months)
- Urine or serum pregnancy test for all females of child-bearing potential
- Chemistry panel, liver function tests, and thyroid stimulating hormone

DSS-2\_05-Oct-2021 

601

602

603

604

605

606 607

608

609

610

611

615

616

618

621

622

623 624

625

626

627

628

629

630

631

• Diabetes Management Information: participant's typical insulin dosing routine including average total daily insulin use (calculated over 1 week), basal rates, carbohydrate ratio(s), and correction factor(s)

Screening procedures will last approximately 2 hours. Once all results of the screening evaluations are available, a decision will be made to determine the participant's eligibility for the study or if one or more part of the screening will have to be repeated. If at the first screening or repeat screening an exclusionary condition is identified, the participant will be excluded from participation with follow up and referred to their primary care physician as needed. The study physician may elect to rescreen participants and collect additional laboratory values if their clinical situation changes.

#### 3.3. Participant Inclusion Criteria

- The participants must meet all of the following inclusion criteria in order to be eligible to participate in the study.
- Age 18 years and older
  - Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least one year
- HbA1c 6.0-11.0%, inclusive
  - Demonstration of proper mental status and cognition for the study
- If on a non-insulin hyperglycemic therapy, stability on that therapy for the prior 3 months and willingness not to alter the therapy for the study duration.
  - For females, not currently known to be pregnant
  - If female and sexually active, must agree to use a highly effective form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study. Also, subjects who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
  - Subjects must have Internet access and a computer system that meets the requirements for uploading the study equipment and ability to participate in video conferencing.
  - Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol

DSS-2\_05-Oct-2021 

663

| 632 | 3.4. | Participant Exclusion Criteria | |
|---|---|---|---|
| 633<br>634 | The pa | rticipant must not have any exclusion criteria in order to be eligible to participate in the | |
| 635 | • | NPH (n | eutral protamine hagedorn) insulin |
| 636<br>637 | • | Use of any medication that at the discretion of the investigator is deemed to interfere with the trial. | |
| 638 | • | Current treatment of a primary seizure disorder | |
| 639<br>640 | • | Coronary artery disease or heart failure, unless written clearance is received from a cardiologist. | |
| 641 | • | Hemophilia or any other bleeding disorder | |
| 642<br>643 | • | A known medical condition, which in the opinion of the investigator or designee, would put the participant or study at risk such as the following examples: | |
| 644 | | 0 | Inpatient psychiatric treatment in the past 6 months |
| 645 | | 0 | Presence of a known adrenal disorder |
| 646<br>647 | | | Abnormal liver function test results (Transaminase >3 times the upper limit of normal) |
| 648 | | 0 | Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2). |
| 649 | | 0 | Active gastroparesis requiring medical therapy |
| 650 | | 0 | Uncontrolled thyroid disease (TSH undetectable or >10 mIU/L). |
| 651 | | 0 | Abuse of alcohol or recreational drugs |
| 652<br>653 | | | Infectious process not anticipated to be resolved prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis, deep tissue infection). |
| 654<br>655 | | | Uncontrolled arterial hypertension (Resting diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg). |
| 656<br>657<br>658 | | | Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy or VEGF inhibitor injections) in the past 12 months. |
| 659<br>660<br>661 | • | A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol. | |
| 662 | • | Not fan | niliar with smart phone technology |

DSS-2\_05-Oct-2021 

• Current use of the following drugs and supplements:

688

689

664 Oral steroids 665 Any other medication that the investigator believes is a contraindication to the subject's participation 666 667 Participation in another pharmaceutical or device trial at the time of enrollment or during 668 the study. 669 Screening procedures will last approximately 2 hours. Once all results of the screening 670 evaluations are available, a decision will be made to determine the participant's eligibility for the 671 study or if one or more parts of the screening will have to be repeated. If at the first screening or 672 repeat screening an exclusionary condition is identified, the participant will be excluded from 673 participation with follow up and referred to their primary care physician as needed. The study 674 physician may elect to rescreen participants and collect additional laboratory values if their 675 clinical situation changes. 676 3.5. **Post-screening assessments** 677 If the subject is deemed eligible to participate in the study, the subject will elect to use either 678 continuous subcutaneous insulin infusion (CSII) or MDI therapy for the duration of the study, no 679 changes are allowed during the study. Furthermore, the participant will elect to use 680 carbohydrates counting or not for the computation of the meal bolus, this choice will apply to 681 the entire study. 682 Participants will then go through a baseline psycho-behavioral assessment. The following questionnaires will be completed: 683 Diabetes Specific Personality Questionnaire 684 685 **ABACUS** Diabetes Locus of Control 686 687 • Confidence in Diabetes Self-Care Scale

Clarke's Hypoglycemia Awareness Scale Participant Inclusion Criteria

Demographic Data Survey (screening visit only)

DSS-2\_05-Oct-2021 

# **Chapter 4** Training Visit

- 691 Participants may use CSII or multiple daily insulin (MDI) injection therapy for their diabetes
- 692 management. Participants will be asked to maintain this treatment throughout the study. In the
- 693 event that MDI participants elects to change to CSII therapy (see section 3.5), the run-in period
- 694 will include a period of insulin stabilization for up to 6 weeks. The study physician may elect to
- 695 extend this time frame if additional time would be beneficial to the participant.
- 696 If participants intend on identifying carbohydrate counting (carbohydrate ratio, insulin sensitivity
- factor and glucose goal) at mealtime, they will be asked to continue to provide this information
- 698 throughout the study.

690

700

#### 699 4.1. Visit 2 - Study Equipment

#### 4.1.1. Study Continuous Glucose Monitor Training

- 701 A Dexcom G6 CGM will be provided to all participants at the training session. The participants
- 702 will be provided with CGM equipment and instructed to use the study CGM on a daily basis. If
- the participant has prior use of the CGM, re-training will be specific to the individual. The study
- team may elect to have less frequent CGM users watch the Dexcom online training videos
- 705 (https://www.dexcom.com/training-videos) to assist in the training session. Study staff training
- 706 may include review of study CGM in real-time to make management decisions and how to review
- 707 the data after an upload for retrospective review. Study staff will specifically identify how alarms
- are set using the app and the frequency that these alarms will repeat when enabled.
- 709 The participants personal CGM will be discontinued. The participants will be observed placing the
- 710 sensor and will learn/review how to access the CGM trace. The participants will be asked to
- 711 perform fingerstick blood glucose measurements (if needed) in accordance with the labeling of
- 712 the study CGM device.
- 713 An electronic copy of the CGM user's guide will be provided for the participants to take home.
- 714 The study team will be sure that the participants will leave the clinic knowing how to properly
- 715 use the CGM.
- 716 Upon request, the study team will provide a Dexcom receiver to allow participants to share their
- 717 CGM data with their personal care providers.

#### 718 4.1.2. Study Pump (Tandem t:AP) Training (CSII participants)

- 719 Eligible participants will be fully instructed on the study insulin pump. A qualified staff member
- 720 will conduct the training and discuss particular differences from the home pump in important
- aspects such as calculation of insulin on board and correction boluses.

DSS-2\_05-Oct-2021 

- 722 Additional training topics are not limited to but may include: infusion site initiation,
- 723 cartridge/priming procedures, setting up the pump, charging the pump, navigation through
- menus, bolus procedures including stopping a bolus, etc.
- 725 The study pump will be programmed with the subject's usual basal rates and pump parameters.
- 726 The study team will assist the subject in study pump infusion site initiation and will assist the
- 727 subject on starting the study pump.
- 728 The subject's personal pump will be removed.
- 729 The subject will be supervised with the study pump during at least one meal or snack bolus to
- 730 ensure subject understanding of the pump features.
- 731 The subject will be encouraged to review the literature provided with the pump and infusion sets
- 732 after the training is completed.

#### 733 **4.1.3. DiAs Training**

- Prior to initial use, the DiAs will be initialized by a study team member with the participant's
- 735 individual insulin dosing parameters, including carbohydrate ratio, insulin sensitivity factor and
- 736 basal insulin doses. If applicable, the study team will confirm the carbohydrate counting
- 737 parameters entered in the system with the study physician.
- 738 Qualified study team members will train the subject in performing specific tasks including the
- 739 following:

740

741

742

743

744

745746

747

750

751752

753

- How to view the CGM information including the most recent CGM value, trend arrow, and CGM graph. Low and high threshold alerts will be set. The patient may choose the threshold alert values, but the low alert may not be set to <70 mg/dL and the high alert may not exceed 300 mg/dL.
- How to connect the CGM transmitter to DiAs as well as troubleshooting techniques for reconnecting. If the CGM values are not available, the subject will be asked to perform fingerstick BG measurements for insulin dosing and treatment management.
- How to start and stop a sensor session with the DiAs APP.
- [for CSII participants] How to connect the pump to DiAs and troubleshooting steps for reconnection.
  - [For MDI participants] How to retroactively inform the system of past insulin doses
  - How to activate the "meal" screen of the DiAs system any time meal insulin or additional correction insulin is desired. And how to use the selected bolus calculator (different if counting carbohydrates or not, see section 3.5).

DSS-2\_05-Oct-2021 

- How to inform the system of hypoglycemia treatment via a "hypoglycemia treatment"
   button on the DiAs user interface after glucose is consumed that is not accompanied by
   an insulin bolus.
- What to do when exercising while using the system and how to use a temporary basal rate.
- How to accept DiAs mode changes sent remotely by the study team.
- 760 DiAs instructions will be provided in the study training manual.

#### 761 **4.1.4. Ketone Meter Training**

- Subjects will be provided with a study blood ketone meter, test strips, and standard control
- solution to perform QC testing per manufacturer guidelines. QC will be completed prior to subject
- 764 receiving the study ketone meter. Only meters that read within the target range at two
- concentrations per manufacturer labeling will be used in the study. The subject will be instructed
- to contact study staff for a replacement of the meter, test strips, and control solution if a meter
- 767 fails QC testing at home.
- 768 Subjects will be instructed to perform blood ketone testing per the Glycemic Treatment
- 769 Guidelines located in the study training manual.

#### 770 4.2. Ecological Momentary Assessment Training

- 771 After randomization, all participants will be trained on how to access and complete EMAs from
- 772 their study phone, how to postpone alerts, and enter a voluntary diary. Participants will be
- informed when the EMAs are scheduled during each phase of the trial.

#### 774 4.3. Glucagon Emergency Kit

- 775 A home glucagon emergency kit will be required. Participants who currently do not have one will
- be given a prescription for the glucagon emergency kit.

DSS-2\_05-Oct-2021 
## **Chapter 5** Study Procedures

#### 778 **5.1. Study Contacts**

777

#### 779 **5.1.1.** Study Support

- 780 Participants will also receive study staff contact information to ask any questions they may have
- during the study. Additionally, participants will be provided with study contact information for
- technical support with DiAs System, the study insulin pump and the study CGM. The participant
- 783 will be asked to call the study team at any time during the study for any health-related issues
- 784 (adverse events), including hypoglycemia <54 mg/dL, frequent highs >300 mg/dL, or ketones ≥3.0
- 785 mmol/L. The participant may use the study pump and study CGM during periods of DiAs
- 786 disconnections or technical difficulties.

#### 787 **5.1.2.** Web Conferencing

- 788 Study visits may be completed using HIPAA compliant web conference tool. The study team will
- provide the participant with the meeting information in advance of the appointment.

## 790 5.2. Sensor-Augmented Mode (SAM) Run-in Period

#### 791 **5.2.1. CGM** use

- 792 Once all training activities are completed, the participant will be given adequate supplies to
- 793 complete the Run-in home use of the DiAs system in SAM.
- 794 Participants will complete a minimum of 14 days (if CGM use within the preceding 3 months) or
- 795 4 weeks (if no CGM use within the preceding 3 months) of home use of the DiAs system in SAM.
- 796 The study physician may request an additional run-in period of 2 weeks.
- 797 The participant will be informed that in order to be eligible for the study, the DiAs system in SAM
- must be used on a minimum of 11 out of 14 days for CGM users or 22 out of 28 days CGM
- 799 nonusers.
- An appointment for Visit 3 will be scheduled.

#### 801 **5.2.2. Questionnaires**

- Participants will be sent the following questionnaires on the final week of the Run-in Period and
- will be asked to complete them within 1 week:
- T1-Diabetes Distress Scale
- Hypoglycemia Fear Survey

DSS-2\_05-Oct-2021 

Hyperglycemia Avoidance Scale

806

807

5.3.

808 The participant may complete this visit via web conferencing and/or at the study site. 809 5.3.1. **Eligibility Assessment** The CGM and insulin data will be reviewed to assess whether the subject has used the DiAs 810 system in SAM on at least 11 out of 14 days for CGM users or 22 out of 28 days for non-CGM 811 812 users. Subjects who are unable to meet the CGM and DiAs compliance requirement will be withdrawn from the study, unless the investigator believes that there were extenuating 813 circumstances that prevented successful completion. In such cases, the investigator may ask the 814 participant to repeat this eligibility assessment. 815 816 5.3.2. **Adverse Event Assessment** 817 The participant will be asked about any of adverse events, adverse device effects, and device issues since the last visit. The participant will also be asked if there were any low BGs <54 mg/dL, 818 819 high BGs >300 mg/dL, or ketones ≥3.0 mmol/L since the last visit. Participants will be encouraged 820 to contact the study team between visits as needed (i.e. report adverse events in real-time).

Visit 3 – Eligibility Assessment, Randomization and Training

DSS-2\_05-Oct-2021 

821

## Chapter 6 Study Procedures - Escalation

- 822 **6.1.1.** Randomization to Escalation
- 823 Eligible subjects will be randomized to therapy escalation (SAM $\rightarrow$ PF $\rightarrow$ DSS).
- A baseline Hemoglobin A1C will be collected. The participant will receive a mode change for
- Phase 1 according to the randomization scheme.
- 826 **6.2. Sensor Augmented Mode**
- 827 Participants randomized to escalation will have any questions answered about continuing use of
- 828 the DiAs system in SAM.
- 829 **6.2.1. SAM EMA Surveys**
- Over the course of 2-3 days every two weeks of Phase 2, the participant will be asked to complete
- a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per
- 832 participant during each Phase.
- 833 **6.2.2. Phase 1 Initiation Questionnaires**
- Participants randomized to escalation will complete the following questionnaires:
- Pittsburgh Sleep Quality Index
- 836 Once all training activities are completed, the participant will be given adequate supplies and
- study devices to last until the subsequent clinic visit. An appointment for Visit 4 will be scheduled
- 838 6.3. Home Use of DiAs in Phase 1 Mode
- The participant will complete a minimum of 8 weeks of DiAs use in Phase 1 Mode at home. During
- the course of Phase 1, participants will complete EMA surveys and post-phase questionnaires.
- 841 **6.3.1. Phase 1 EMA Surveys**
- Over the course of 2-3 days every two weeks of Phase 1, the participant will be asked to complete
- a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per
- 844 participant during each Phase.
- 845 **6.3.2.** Post-Phase 1 Questionnaires Week 7
- Participants randomized to escalation will be sent the following questionnaires on week 7 (day
- 42 of Phase 1) and will be asked to complete them within 1 week:
- Pittsburgh Sleep Quality Index

DSS-2\_05-Oct-2021 

878

• INSPIRE (revised for DSS)

| 349 | Hyperglycemia Avoidance Scale |
|---|---|
| 50 | 5.3.3. Post-Phase 1 Questionnaires Week 8 |
| 351<br>352 | Participants randomized to escalation will sent the following questionnaires on week 8 (day 4 of Phase 1) and will be asked to complete them within 1 week: |
| 353 | Confidence in Diabetes Self-Care Scale |
| 854 | T1-Diabetes Distress Scale |
| 355 | Hypoglycemia Fear Survey |
| 356 | 5.4. Visit 4 – Phase 2 Initiation |
| 857<br>858<br>859<br>860<br>861 | All participants in each randomization scheme use PF in Phase 2. Phase 2 initiation may be conducted either via web conference or an office visit. The participant will remotely receive mode change for Phase 2. Study staff will review the features of the Personalized Feedback (PF mode and answer any questions. Participant will have a blood/urine pregnancy test that must be negative in order to continue to participate in this study. |
| 362 | 6.4.1. Training on Phase 2 DiAs Mode |
| 363<br>364<br>365<br>366<br>367<br>368<br>369<br>370<br>371<br>372<br>373 | <ul> <li>Tracking of estimated HbA1c: When properly calibrated, eA1c is within 0.3% of reference HbA1c on average, and within 1% of HbA1c &gt;95% of the time.</li> <li>Hypoglycemia Risk Indicator: Provides an indication of the current risk for hypoglycemia.</li> <li>Insulin Sensitivity Profile &amp; Indicator: Tracks changes in insulin sensitivity (SI) and creates daily and monthly SI profiles.</li> <li>Insulin on Board: Tracks active insulin to avoid insulin stacking using a common 4-6 hou action curve.</li> <li>Personalized weekly feedback. Provides advice to the user on what went well in terms of glycemic control and system use in the past week and what may be a good thing to focus on for the following week.</li> </ul> |
| 875 | 5.4.2. Phase 2 Initiation Questionnaires |
| 876 | Participants randomized to escalation will complete the following questionnaires: |
| 377 | Technology Expectations (burdens subscale only) |

DSS-2\_05-Oct-2021 

905

906

Hyperglycemia Avoidance Scale

• Confidence in Diabetes Self-Care Scale

#### 879 6.4.3. Adverse Event Assessment 880 The participant will be asked about any of adverse events, adverse device effects, and device 881 issues since the last visit. The participant will also be asked if there were any low BGs <54 mg/dL, 882 high BGs >300 mg/dL, or ketones ≥3.0 mmol/L since the last visit. 883 Once all training activities are completed, the participant will be given adequate supplies and 884 study devices to last until the subsequent clinic visit. An appointment for Visit 5 will be scheduled. 885 Participants will be encouraged to contact the study team between visits as needed (i.e. report 886 adverse events in real-time). Home Use of DiAs in Phase 2 Mode 887 6.5. 888 The participant will complete a minimum of 8 weeks of DiAs use in Phase 2 Mode at home. 889 During the course of Phase 2, participants will complete EMA surveys and post-phase 890 questionnaires. 891 6.5.1. **Phase 2 EMA Surveys** Over the course of 2-3 days every two weeks of Phase 2, the participant will be asked to complete 892 893 a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per participant during each Phase. 894 895 Post-Phase 2 Questionnaires Week 7 6.5.2. 896 All participants will be sent the following questionnaires on week 7 (day 42 of Phase 2) and will 897 be asked to complete them within 1 week: 898 Technology Acceptance (burdens subscale only) 899 Pittsburgh Sleep Quality Index 900 T1-Diabetes Distress Scale Post-Phase 2 Questionnaires Week 8 901 6.5.3. 902 All participants will be sent the following questionnaires on week 8 (day 49 of Phase 2) and will 903 be asked to complete them within 1 week: 904 Hypoglycemia Fear Survey

DSS-2\_05-Oct-2021 

#### 907 **6.6. Visit 5 – Phase 3 Initiation**

- 908 The participant will begin Phase 3 according to the randomization scheme either via web
- conference or an office visit. The participant will remotely receive a mode change for Phase 3.
- 910 Study staff will review the features of the Phase 3 system and answer any questions. Participant
- 911 will have a blood/urine pregnancy test that must be negative in order to continue to participate
- 912 in this study.

920

921

922

923

924

925

926

927

928

#### 913 **6.6.1.** Training on Phase 3 DiAs Mode

- Participants randomized to escalation will be trained to use DiAs in DSS mode, including the following features:
- Exercise Advice: An advisory module that ensures safety of mild to moderate exercise by predicting whether an exercise bout is likely to result in hypoglycemia and providing a graded carbohydrate supplementation strategy and possible reduction in insulin advice.
  - **Bedtime Advice:** Gauges overnight hypoglycemia risk and provides bedtime carbohydrate advice.
  - Smart Bolus Calculator: An advanced bolus calculator capable of accounting for several factors such as exercise (activity on board), metabolic characteristics (correction based on 45 min predicted glucose to account for insulin delays) and SI fluctuations (insulin sensitivity tracker).
  - Treatment Parameter Optimization: An optimization routine that analyzes the previous 30 days of CGM, insulin, and meal data to provide updated insulin treatment parameters (CR, CF, and basal rate) to minimize glycemic risk.

#### 929 **6.6.2.** Phase 3 Initiation Questionnaires

- 930 Participants randomized to escalation will complete the following questionnaires:
- Technology Expectations (burdens subscale only)
- INSPIRE (revised for DSS)
- Diabetes Locus of Control

#### 934 **6.6.3.** Adverse Event Assessment

- The participant will be asked about any of adverse events, adverse device effects, and device
- 936 issues since the last visit. The participant will also be asked if there were any low BGs <54 mg/dL,
- 937 high BGs >300 mg/dL, or ketones ≥3.0 mmol/L since the last visit. Participants will be encouraged
- to contact the study team between visits as needed (i.e. report adverse events in real-time).

DSS-2\_05-Oct-2021 

967

ABACUS

| 6.7. | Home Use of DiAs in Phase 3 Mode |
|---|---|
| • | orticipant will complete a minimum of 8 weeks of Phase 3 at home. During the course of 3, participants will complete EMA surveys and post-phase questionnaires. |
| 6.7.1. | Phase 3 EMA Surveys |
| a "Dai | he course of 2-3 days every two weeks of Phase 3, the participant will be asked to complete<br>y Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per<br>pant during each Phase. |
| 6.7.2. | Post-Phase 3 Questionnaires Week 7 |
| | pants randomized to escalation will be sent the following questionnaires on week 7 (day Phase 1) and will be asked to complete them within 1 week: |
| | Technology Acceptance (burdens subscale only) |
| | Pittsburgh Sleep Quality Index. |
| | • T1-Diabetes Distress Scale |
| 6.7.3. | Post-Phase 3 Questionnaires Week 8 |
| | pants randomized to escalation will sent the following questionnaires on week 8 (day $49$ se 3) and will be asked to complete them within 1 week: |
| | Hypoglycemia Fear Survey |
| | Hyperglycemia Avoidance Scale |
| | Confidence in Diabetes Self-Care Scale |
| 6.8. | Visit 6 - Study Exit |
| Partici | pants will participate in a Study Exit visit either via web conference or an office visit pants will return to their standard diabetes care using their personal equipment. The study will be available to answer questions about insulin parameters. |
| study, | orticipant will be asked to return all investigational study devices (e.g. study insulin pump<br>CGM, study phone, other associated supplies) either via mail or at an office visit<br>pants may keep the study glucometer and ketone meter. |
| 6.8.1. | Study Exit Questionnaires |
| Partici | pants randomized to escalation will complete the following questionnaires: |

DSS-2\_05-Oct-2021 

| 968 | • | INSPIRE (revised for DSS) |
|---|---|---|
| 969 | • | Diabetes Locus of Control |
| 970 | 6.8.2. | Adverse Event Assessment |
| 971<br>972<br>973 | issues | rticipant will be asked about any of adverse events, adverse device effects, and device since the last visit. The participant will also be asked if there were any low BGs <54 mg/dLGs >300 mg/dL, or ketones ≥3.0 mmol/L since the last visit. |
| 974 | 6.9. | Post Study Check-In Visit (Visit 7) |
| 975<br>976 | • • | kimately 48 hours after the home use of the equipment, the study team will contact the pant via phone/email/text to assess: |
| 977 | • | Adverse events, adverse device effects, and device issues |
| 978 | • | Blood glucose values <60 mg/dL and >300 mg/dL |

DSS-2\_05-Oct-2021 

979

987

988

989

990

991

992993

994

995

996

997

998

## Chapter 7 Study Procedures – De-Escalation

- 980 7.1. Randomization to De-Escalation
- 981 Eligible subjects will be randomized to therapy de-escalation (DSS $\rightarrow$ PF $\rightarrow$ SAM).
- 982 A baseline Hemoglobin A1C will be collected.
- The participant will receive a mode change for Phase 1 according to the randomization scheme.
- 984 7.2. Training on Phase 1 DiAs Mode
- Participants randomized to de-escalation will be trained to use DiAs in DSS mode, including the following features:
  - Exercise Advice: An advisory module that ensures safety of mild to moderate exercise by
    predicting whether an exercise bout is likely to result in hypoglycemia and providing a
    graded carbohydrate supplementation strategy and possible reduction in insulin advice.
  - Bedtime Advice: Gauges overnight hypoglycemia risk and provides bedtime carbohydrate advice.
    - Smart Bolus Calculator: An advanced bolus calculator capable of accounting for several factors such as exercise (activity on board), metabolic characteristics (correction based on 45 min predicted glucose to account for insulin delays) and SI fluctuations (insulin sensitivity tracker).
    - Treatment Parameter Optimization: An optimization routine that analyzes the previous 30 days of CGM, insulin, and meal data to provide updated insulin treatment parameters (CR, CF, and basal rate) to minimize glycemic risk.
- 999 **7.2.1.** Phase 1 EMA Surveys
- Over the course of 2-3 days every two weeks of Phase 2, the participant will be asked to complete
- a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per
- 1002 participant during each Phase.
- 1003 7.2.2. Phase 1 Initiation Questionnaires
- 1004 Participants randomized to de-escalation will complete the following questionnaires:
- 1005 Pittsburgh Sleep Quality Index
- Technology Expectations (burdens subscale only)
- INSPIRE (revised for DSS)
- Once all training activities are completed, the participant will be given adequate supplies and study devices to last until the subsequent clinic visit. An appointment for Visit 4 will be scheduled.

DSS-2\_05-Oct-2021 

Home Use of DiAs in Phase 1 Mode

7.3.

1010

10351036

1037

1038

| The participant will complete a minimum of 8 weeks of DiAs use in Phase 1 Mode at home. During the course of Phase 1, participants will complete EMA surveys and post-phase questionnaires. |
|---|
| 7.3.1. Phase 1 EMA Surveys |
| Over the course of 2-3 days every two weeks of Phase 1, the participant will be asked to complete a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per participant during each Phase. |
| 7.3.2. Post-Phase 1 Questionnaires Week 7 |
| Participants randomized to de-escalation will be sent the following questionnaires on week 7 (day 42 of Phase 1) and will be asked to complete them within 1 week: |
| Technology Acceptance (burdens subscale only) |
| Pittsburgh Sleep Quality Index |
| T1-Diabetes Distress Scale |
| 7.3.3. Post-Phase 1 Questionnaires Week 8 |
| Participants randomized to de-escalation will be sent the following questionnaires on week 8 (day 49 of Phase 1) and will be asked to complete them within 1 week: |
| Hypoglycemia Fear Survey |
| Hyperglycemia Avoidance Scale |
| Confidence in Diabetes Self-Care Scale |
| 7.4. Visit 4 – Phase 2 Initiation |
| All participants in each randomization scheme use PF in Phase 2. Phase 2 initiation may be conducted either via web conference or an office visit. The participant will remotely receive a mode change for Phase 2. Study staff will review the features of the Personalized Feedback (PF) mode and answer any questions. |
| 7.4.1. Training on Phase 2 DiAs Mode |

DSS-2\_05-Oct-2021 

The participant will be trained on the following features of the Personalized Feedback System:

HbA1c on average, and within 1% of HbA1c >95% of the time.

• Tracking of estimated HbA1c: When properly calibrated, eA1c is within 0.3% of reference

• **Hypoglycemia Risk Indicator:** Provides an indication of the current risk for hypoglycemia.

- Insulin Sensitivity Profile & Indicator: Tracks changes in insulin sensitivity (SI) and creates
   daily and monthly SI profiles.
- **Insulin on Board:** Tracks active insulin to avoid insulin stacking using a common 4-6 hour action curve.
  - **Personalized weekly feedback.** Provides advice to the user on what went well in terms of glycemic control and system use in the past week and what may be a good thing to focus on for the following week.

#### 1046 **7.4.2. Phase 2 Initiation Questionnaires**

- 1047 Participants randomized to de-escalation will complete the following questionnaires:
- Technology Expectations (burdens subscale only)
- INSPIRE (revised for DSS)
- 1050 Diabetes Locus of Control

#### 1051 **7.4.3. AE Assessment**

1043

1044

1045

- The participant will be asked about any of adverse events, adverse device effects, and device
- issues since the last visit. The participant will also be asked if there were any low BGs <54 mg/dL,
- high BGs >300 mg/dL, or ketones ≥3.0 mmol/L since the last visit.
- Once all training activities are completed, the participant will be given adequate supplies and
- study devices to last until the subsequent clinic visit. An appointment for Visit 5 will be scheduled.
- 1057 7.5. Home Use of DiAs in Phase 2 Mode
- The participant will complete a minimum of 8 weeks of DiAs use in Phase 2 Mode at home.
- 1059 During the course of Phase 2, participants will complete EMA surveys and post-phase
- 1060 questionnaires.

#### 1061 **7.5.1.** Phase 2 EMA Surveys

- Over the course of 2-3 days every two weeks of Phase 2, the participant will be asked to complete
- a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per
- 1064 participant during each Phase.

#### 1065 7.5.2. Post-Phase 2 Questionnaires Week 7

- 1066 All participants will be sent the following questionnaires on week 7 (day 42 of Phase 2) and will
- be asked to complete them within 1 week:
- Technology Acceptance (burdens subscale only)

DSS-2\_05-Oct-2021 

1097

1098

| .069 | Pittsburgh Sleep Quality Index |
|---|---|
| .070 | T1-Diabetes Distress Scale |
| .071 | 7.5.3. Post-Phase 2 Questionnaires Week 8 |
| .072<br>.073 | All participants will be sent the following questionnaires on week 8 (day 49 of Phase 2) and will be asked to complete them within 1 week: |
| .074 | Hypoglycemia Fear Survey |
| .075 | Hyperglycemia Avoidance Scale |
| .076 | Confidence in Diabetes Self-Care Scale |
| .077 | 7.6. Visit 5 – Phase 3 Initiation |
| .078<br>.079<br>.080 | The participant will begin Phase 3 according to the randomization scheme either via web conference or an office visit. The participant will remotely receive a mode change for Phase 3. Study staff will review the features of the Phase 3 system and answer any questions. |
| .081 | 7.6.1. Training on Phase 3 DiAs Mode |
| .082<br>.083 | Participants randomized to de-escalation will have any questions answered about resuming use of the DiAs system in SAM. |
| .084 | 7.6.2. Phase 3 Initiation Questionnaires |
| .085<br>.086<br>.087 | Participants randomized to de-escalation will complete the following questionnaires: • INSPIRE (revised for DSS) • Diabetes Locus of Control |
| .088 | 7.6.3. Adverse Event Assessment |
| .089<br>.090<br>.091 | The participant will be asked about any of adverse events, adverse device effects, and device issues since the last visit. The participant will also be asked if there were any low BGs <54 mg/dL, high BGs >300 mg/dL, or ketones ≥3.0 mmol/L since the last visit. |
| .092<br>.093<br>.094<br>.095 | Once all training activities are completed, the participant will be given adequate supplies and study devices to last until the subsequent clinic visit. An appointment for Visit 6 will be scheduled. Participants will be encouraged to contact the study team between visits as needed (i.e. report adverse events in real-time). |
| .096 | 7.7. Home Use of DiAs in Phase 3 Mode |

DSS-2\_05-Oct-2021 

The participant will complete a minimum of 8 weeks of Phase 3 at home. During the course of

Phase 3, participants will complete EMA surveys and post-phase questionnaires.

DSS-2\_05-Oct-2021 

| 1128 | 7.9. Post Study Check-In Visit (Visit 7) |
|---|---|
| 1129 | Approximately 48 hours after the home use of the equipment, the study team will contact the |
| 1130 | participant via phone/email/text to assess: |
| 1131 | Adverse events, adverse device effects, and device issues |
| 1132 | <ul> <li>Blood glucose values &lt;60 mg/dL and &gt;300 mg/dL</li> </ul> |

DSS-2\_05-Oct-2021 

# 1133 Chapter 8 Testing Procedures

#### 1134 8.1. Laboratory / Point of Care Testing

- 1135 **8.1.1. HbA1c**
- A blood sample will be obtained at screening to obtain a baseline hemoglobin A1c level.
- HbA1c level may be measured by study team using the DCA2000, a comparable point of
   care device, at time of screening
- Labs may be obtained at a local laboratory (e.g. LabCorp) convenient to the participant.
- Blood test may be obtained within 14 days prior to enrollment may be used for eligibility purposes.
- Sample collected at randomization and end of study will be used for statistical purposes.

#### 1143 **8.1.2.** Comprehensive Metabolic Panel

- A blood sample will be obtained at screening to assess kidney and liver functioning.
- Labs may be obtained at a local laboratory (e.g. LabCorp) convenient to the participant.
- Blood test may be obtained within 14 days prior to enrollment may be used for eligibility
   purposes.

#### 1148 **8.1.3.** Thyroid Stimulating Hormone

- A blood sample will be obtained at screening to assess thyroid function.
- Labs may be obtained at a local laboratory (e.g. LabCorp) convenient to the participant.
- Blood test may be obtained within 14 days prior to enrollment may be used for eligibility purposes.

#### 1153 **8.1.4. Pregnancy Test**

- 1154 A blood/urine pregnancy test will be required for women of childbearing potential at the
- screening visit, and between each phase . Tests must be negative to participate in the study.

DSS-2\_05-Oct-2021 

## **Chapter 9** Questionnaires & Ecological Momentary Analysis

#### 9.1. Diabetes Specific Personality Questionnaire

- 1158 The Diabetes Specific Personality Questionnaire is based on the original Six Factor Personality
- 1159 Questionnaire [81], a well-validated measure that was adapted for the diabetes-specific version
- of the questionnaire. The Six Factor Personality Questionnaire is a measure of six personality
- dimensions each consisting of three facet scales, measured by 108 Likert items. The Six Factor
- 1162 Personality Questionnaire facet scales are organized in terms of six factor scales. The Diabetes
- 1163 Specific Personality Questionnaire assesses three personality factors conscientiousness,
- obsessive-compulsiveness, and openness. In this study, the Diabetes Specific Personality
- 1165 Questionnaire is used to explore whether personality type is associated with willingness and/or
- ability to effectively engage with the DSS. Administration time is approximately 15 minutes.

#### 1167 **9.2. ABACUS**

1156

1157

1175

1182

- 1168 This is a structured interview used to provide a very brief assessment of carbohydrate counting
- and diabetes self-management skills important to effective engagement consisting of a series of
- 1170 25 questions assessing health literacy and health numeracy in people with T1DM [84].. The
- interviewer evaluates the subject answer to each question on a scale ranging from 1 (No
- competency) to 3 (Full competency); the sum yields to a total score. The higher the score, the
- 1173 higher the levels of health literacy and numeracy of the subject. Administration time is
- approximately 10-20 minutes.

#### 9.3. Diabetes Locus of Control

- 1176 This questionnaire [85] was developed for use on adults (18-80 y.o.) The scale consists of 18 items
- 1177 measuring the individual's personal beliefs about their control over their diabetes management
- and outcome: 6 items measuring internal locus of control, 6 items measuring powerful others
- locus of control, and 6 items measuring chance locus of control. A 6-point Likert-type scale is used
- in which 0 indicates 'strongly disagree with the statement' and 5 indicates 'strongly agree with
- the statement.' Administration time is approximately 5 minutes.

#### 9.4. Confidence in Diabetes Self-Care Scale

- 1183 This is a short 20-item self-report questionnaire assessing self-efficacy, the perceived ability to
- 1184 perform diabetes self-care tasks, in patients with T1DM [87]. Items are constructed to cover all
- domains of self-care as well as social skills. Each item is preceded by, "I believe I can..." with the
- strength of this belief rated on a 5-point Likert scale ranging from 1 ("No, I am sure I cannot") to
- 1187 5 ("Yes, I am sure I can"). Administration time is approximately 10 minutes.

DSS-2\_05-Oct-2021 

1188

1201

1212

#### 9.5. Clarke's Hypoglycemia Awareness Scale

- 1189 The scale comprises eight questions characterizing the participant's level of hypoglycemia
- awareness, as well as risk for exposure to episodes of moderate and severe hypoglycemia [88].
- 1191 It also examines the glycemic threshold for symptomatic responses to hypoglycemia. A score of
- four or more on a scale of 0 to 7 implies impaired awareness of hypoglycemia. Administration
- time is approximately 5 minutes.

#### 1194 9.6. The Diabetes Distress Scale

- 1195 This is a measure that reflects diabetes-specific quality of life and emotional well-being [90]. The
- Diabetes Distress Scale is a measure of diabetes-related distress over a number of domains (e.g.
- diabetes management regimen, interpersonal distress) and consists of a scale of 17 items. These
- include items from each of four domains central to diabetes-related emotional distress. Patients
- rate the degree to which each item is currently problematic for them on a 6-point Likert scale,
- from 1 (no problem) to 6 (serious problem). Administration time is approximately 5 minutes.

#### 9.7. Hypoglycemia Fear Survey

- 1202 This guestionnaire will be used to determine if the PF and DSS is associated with reduced fear of
- 1203 hypoglycemia. The Hypoglycemia Fear Survey-II [91] was developed to measure behaviors and
- worries related to fear of hypoglycemia in adults with T1DM. It is composed of 2 subscales, the
- 1205 Behavior and Worry. Behavior items describe behaviors in which patients may engage to avoid
- 1206 hypoglycemic episodes and/or their negative consequences (e.g., keeping blood glucose levels
- higher, making sure other people are around, and limiting exercise or physical activity). Worry
- 1208 items describe specific concerns that patients may have about their hypoglycemic episodes (e.g.,
- being alone, episodes occurring during sleep, or having an accident). Items are rated on a 5-point
- 1210 Likert scale (0=never, 4=always), with higher scores indicating higher fear of hypoglycemia.
- 1211 Administration time is approximately 10 minutes.

#### 9.8. Hyperglycemia Avoidance Scale

- 1213 This measure is used to assess the extent of potentially problematic avoidant attitudes and
- 1214 behaviors in people with T1DM [91]. The Hypoglycemia Avoidance Scale reliably quantifies
- affective and behavioral aspects of hyperglycemia avoidance and is used to assess the extent of
- 1216 potentially problematic avoidant attitudes and behaviors regarding hyperglycemia in people with
- 1217 T1DM. It has 24 items plus two additional optional items asking about the highest level of daily
- 1218 blood glucose or HbA1c measures the individual would feel comfortable having. Administration
- time is approximately 10 minutes.

DSS-2\_05-Oct-2021 

1220

1237

#### 9.9. Pittsburgh Sleep Quality Index

- 1221 This questionnaire will be used to assess whether the PF and DSS improve sleep quality and
- 1222 quantity. The Pittsburgh Sleep Quality Index [93] is a self-report questionnaire that assesses sleep
- 1223 quality over a 1-month time interval. The measure consists of 19 individual items, creating 7
- 1224 components that produce one global score: the higher the global score, the poorer the sleep
- 1225 quality. Administration time is approximately 5-10 minutes.

#### 1226 9.10. Technology Acceptance and Expectations Survey (burdens subscale only)

- 1227 The Technology Acceptance Surveys [94-95] were developed for an artificial pancreas camp study
- in adolescents. The 38 items in the questionnaire were based on interviews conducted with
- 1229 individuals who had participated in previous artificial pancreas trials about their experience
- regarding the device. It was subsequently adapted to assess these same measures for the PF and
- 1231 DSS. It assesses both positive and negative experiences with PF and DSS, including blood glucose
- management, device burden, and overall satisfaction. Items are rated on a 5-point scale. In this
- study only the burden subscale will be used. The Technology Expectations Survey has the same
- items included on the Technology Acceptance Survey but asks whether the individual expects to
- 1235 experience the various benefits and burdens from use of a device. Administration time is
- 1236 approximately 10 minutes.

#### 9.11. INSPIRE (revised for DSS)

- 1238 This questionnaire will be used to assess patient preferences to support effective onboarding and
- successful continued use of the PF and DSS. The INSPIRE survey was developed to assess various
- aspects of a user's experience regarding automated insulin delivery for both patients and family
- members. The surveys include various topics important to patients with T1DM and their family
- members based upon >200 hours of qualitative interviews and focus groups. It was adapted by
- its developer for use with the PF and DSS. The survey includes 22 items. Response options include
- 1244 a 5-point Likert scale from strongly agree to strongly disagree, along with an N/A option.
- 1245 Administration time is approximately 5 minutes.

#### 1246 9.12. Ecological Momentary Analysis (EMA)

- 1247 In addition to the behavioral data automatically recorded (e.g. insulin dosing, interactions with
- 1248 system), an EMA procedure will be used to track the users' daily experiences of trust in the
- system, emotional well-being, treatment satisfaction, and diabetes-related concerns and burden.
- 1250 Using a brief daily survey, we will capture the dynamic changes in participant experience
- 1251 throughout the day and the associations between users' subjective experience and their
- reactions to/interactions with the PF and DSS devices. This will be the first use of EMA with

decision support systems.

DSS-2\_05-Oct-2021 

| 1254<br>1255<br>1256 | During each treatment condition, over the course of 2-3 days every two weeks, the participant will be asked to complete a "Daily Diary" with 3-5 entries of 3-4 questions each day, for a minimum total of 48 entries per participant during each Phase. |
|---|---|
| 1257<br>1258<br>1259<br>1260 | The DiAs phone will display a text message containing a link to the survey. Surveys will be triggered at fixed times, including a morning survey ~1h after waking up and an end-of-the-day survey around 8-9 PM. Participants will be able to delay (up to 30 min) or skip (up to 2 per day excluding at wake up) surveys for their convenience. |
| 1261<br>1262 | Participants will respond to questions on a 5-point Likert scale (0=Not at All, 4=Extremely). The first Diary for each day will contain two additional items for rating sleep quantity/quality. |
| 1263<br>1264<br>1265 | The Daily Diary questions are shown below and are intended to assess agreement, trust, treatment satisfaction, diabetes burden, self-efficacy, mood valence, energy level, and physical well-being. |
| 1266 | Quality of Life Parameters |
| 1267 | <ul> <li>At this moment, to what extent do you feel</li> </ul> |
| 1268 | Burdened by your diabetes treatment? |
| 1269 | Worried about your blood sugar levels? |
| 1270 | In a positive or good mood? |
| 1271 | Physically well? |
| 1272 | <ul> <li>Sleep Items_(only presented in the first Diary for each day)</li> </ul> |
| 1273 | <ul><li>Was your sleep last night</li></ul> |
| 1274 | Long enough? |
| 1275 | Restful enough? |
| 1276 | <ul> <li>Technology acceptance (only presented in the last Diary for each day)</li> </ul> |
| 1277 | <ul> <li>Today to what extent have you</li> </ul> |
| 1278 | Found (name of program) easy to use? |
| 1279 | Found (name of program) useful? |
| 1280 | Trusted the information given by (name of program)? |
| 1281 | Found (name of program) easy to use? |
| 1282 | Found (name of program) useful? |
| 1283 | Trusted the information given by (name of program)? |

DSS-2\_05-Oct-2021 

## 1284 **9.13.** Questionnaire Schedule

| Timing | Escalation | De-escalation |
|---|---|---|
| Visit 1 – Screening and | Diabetes Specific Pe | rsonality Questionnaire |
| Questionnaires | | SACUS |
| | Diabetes Locus of Control | |
| | | betes Self-Care Scale |
| | Clarke's Hypoglycemia Awareness Scale | |
| Visit 2 – Study Equipment<br>Training | N | lone |
| F: | T1-Diabetes | s Distress Scale |
| Final week of SAM Run-in | Hypoglycen | nia Fear Survey |
| | Hyperglycemia | a Avoidance Scale |
| very a etc. total | Pittsburgh Sleep Quality Index | Pittsburgh Sleep Quality Index |
| Visit 3 Eligibility Assessment, | | Technology Expectations (burdens subscale only) |
| Randomization and Training | | INSPIRE |
| DiAs Use in Phase 1 Mode | EMA Surveys | EMA Surveys |
| | Pittsburgh Sleep Quality | Technology Acceptance (burdens subscale only) |
| Week 7 of DiAs Use in Phase | Hyperglycemia Avoidance Scale | Pittsburgh Sleep Quality Index |
| 1 Mode | _ ·· - <i>'</i> | T1-Diabetes Distress Scale |
| | Confidence in Diabetes Self-Care | Hypoglycemia Fear Survey |
| Week 8 of DiAs Use in Phase | T1-Diabetes Distress Scale | Hyperglycemia Avoidance Scale |
| 1 Mode | Hypoglycemia Fear Survey | Confidence in Diabetes Self-Care Scale |
| | ,608,700 | Sommachise in Bladetes sen Gare soare |
| | Technology Expectations (burdens subscale only) | Technology Expectations (burdens subscale only) |
| Visit 4 Phase 2 Initiation | INSPIRE (revised for DSS) | INSPIRE (revised for DSS) |
| | | Diabetes Locus of Control |
| DiAs Use in Phase 2 Mode | EMA Surveys | EMA Surveys |
| Week 7 of DiAs Use in Phase | Technology Acceptance (burdens subscale only) | |
| 2 Mode | Pittsburgh Sleep Quality Index | |
| 2 Wiode | T1-Diabetes Distress Scale | |
| Week 8 of DiAs Use in Phase | Hypoglycemia Fear | |
| 2 Mode | Hyperglycemia Avoidance Scale | |
| 2 Wiode | Confidence in Diabetes Self-Care Scale | |
| | community in production sent care search | |
| | Technology Expectations (burdens subscale only) | INSPIRE (revised for DSS) |
| Visit 5 Phase 3 Initiation | INSPIRE (revised for DSS) | Diabetes Locus of Control |
| | Diabetes Locus of Control | Diabetes Locus of Collinor |
| | Diabetes Locus of Collifol | |
| DiAs Use in Phase 3 Mode | EMA Surveys | EMA Surveys |
| DIAS USE III FIIASE 3 MODE | | 200 L L C |
| Week 7 of DiAs Use in Phase | Technology Acceptance (burdens subscale only) to | Pittsburgh Sleep Quality Index |
| 3 Mode | assess patients' experienced burdens related to | T1-Diabetes Distress Scale |
| 3 WIOUE | the use of DSS | |
| | Pittsburgh Sleep Quality Index (PSQI) to assess | |
| | whether DSS improves sleep quality and quantity. | |
| | Hypoglycemia Fear Survey | Hypoglycemia Fear Survey |
| Week 8 of DiAs Use in Phase | Hyperglycemia Avoidance | Hyperglycemia Avoidance Scale |
| 3 Mode | Confidence in Diabetes Self-Care Scale | Confidence in Diabetes Self-Care Scale |
| | ABACUS | ABACUS |
| Visit 6 Study Exit | INSPIRE (revised for DSS) | 7.07.000 |
| | Diabetes Locus of Control | |
| | Dianetes Locus di Collilol | |

1285

DSS-2\_05-Oct-2021 

1286

## Chapter 10 Risks, Benefits, and Risk Assessment

#### 1287 10.1. Potential Risks and Benefits of the Investigational Device

- 1288 Risks and Benefits are detailed below. Loss of confidentiality is a potential risk; however, data are
- handled to minimize this risk. Hypoglycemia, hyperglycemia and ketone formation are always a
- risk in participants with T1DM and participants will be monitored for these symptoms.

#### 1291 10.1.1. Venipuncture Risks

- 1292 A hollow needle will be placed in the arm for taking blood samples. Blood draws can cause some
- 1293 common reactions like pain, bruising, or redness at the sampling site. Less common reactions
- include bleeding from the sampling site, formation of a small blood clot or swelling of the vein
- 1295 and surrounding tissues, and fainting.
- 1296 There is the risk of contamination from blood sampling techniques. Hand washing with either
- soap & water or waterless hand sanitizer will be used prior to caring for the study subject. Gloves
- 1298 will be worn during blood sample collection and processing. Medical personnel will continue to
- practice hygiene for the subject's protection (i.e. hand washing, changing gloves frequently,
- 1300 disposing needles properly). Gloves will be removed and hands washed or sanitized prior to
- 1301 leaving and upon return to the subject's room. Soiled linen will be changed to minimize the
- 1302 transfer of pathogenic organisms.

#### 1303 10.1.2. Fingerstick Risks

- About 2 drop of blood will be removed by fingerstick for measuring blood sugars and sometimes
- 1305 HbA1c or other tests. This is a standard method used to obtain blood for routine hospital
- 1306 laboratory tests. Pain is common at the time of lancing. In about 1 in 10 cases, a small amount of
- bleeding under the skin will produce a bruise. A small scar may persist for several weeks. The risk
- of local infection is less than 1 in 1000. This should not be a significant contributor to risks in this
- 1309 study as fingersticks are part of the usual care for people with diabetes.

#### 1310 **10.1.3.** Subcutaneous Catheter Risks

- 1311 Participants using the study pump infusion sets will be at low risk for developing a local skin
- infection at the site of the infusion set placement. Though approved for 3 days of use, if a catheter
- is left under the skin for more than 24 hours it is possible to get an infection where it goes into
- the skin, with swelling, redness and pain. There may be bleeding where the catheter is put in and
- 1315 bleeding under the skin causing a bruise (1 in 10 risk).

DSS-2\_05-Oct-2021 

1316

#### 10.1.4. Sensor Needle Risks

- 1317 Participants using the continuous glucose monitor (CGM) with sensor will be at low risk for
- developing a local skin infection at the site of the sensor needle placement. Though approved for
- 1319 10 days of use, if a catheter is left under the skin for more than 24 hours it is possible to get an
- infection where it goes into the skin, with swelling, redness and pain. There may be bleeding
- where the catheter is put in and bleeding under the skin causing a bruise (1 in 10 risk).
- 1322 Study staff should verbally alert the participant that on rare occasions, the CGM may break and
- leave a small portion of the sensor under the skin that may cause redness, swelling, or pain at
- the insertion site. The participant should be further instructed to notify the study coordinator
- immediately if this occurs.

#### 1326 10.1.5. Risks of Hypoglycemia

- 1327 As with any person having T1DM and using insulin, there is always a risk of having a low blood
- sugar (hypoglycemia). The frequency of hypoglycemia should be no more and possibly less than
- it would be as part of daily living. Symptoms of hypoglycemia can include sweating, jitteriness,
- and not feeling well. Just as at home, there is the possibility of fainting or seizures (convulsions)
- 1331 and subsequently for a few days the participant may not be as aware of symptoms of
- 1332 hypoglycemia. A poorly functioning CGM can periodically display falsely high glucose values,
- which could lead to inappropriate insulin recommendation.

#### 1334 10.1.6. Risks of Hyperglycemia

- 1335 Hyperglycemia and ketonemia could occur if insulin delivery is attenuated or suspended for an
- 1336 extended period or if the pump or infusion set is not working properly. A poorly functioning CGM
- can periodically display falsely high glucose values, which could lead to inappropriate insulin
- 1338 recommendation.

#### 1339 **10.1.7. Risks of Device Reuse**

- 1340 Participant will be informed that FDA or relevant national authorities have approved the insulin
- pump, CGM, glucometer and ketone meter for single use and that by using them among multiple
- patients, bloodborne pathogens (i.e. Hepatitis B) may be spread through the use of multiple
- 1343 users.
- 1344 The study CGM system is labelled for single use only. The sensor (the component of the system
- that enters the skin) will be single use only. The transmitter and receiver may be reused during
- the study after cleaning the device using a hospital-approved cleaning procedure. The transmitter

DSS-2\_05-Oct-2021 

- is attached to the sensor but does not enter the skin and the receiver, if used, is a hand held
- 1348 device.
- 1349 The study insulin pumps are labelled for single-patient use. During the study, this device may be
- reused after adhering to a hospital-approved cleaning procedure. All infusion set equipment will
- be single patient use only (infusion set insertion kits, tubing, cartridges etc.).

#### 1352 **10.1.8.** Other Risks

- 1353 Some participants may develop skin irritation or allergic reactions to the adhesives used to secure
- the CGM, or to secure the insulin infusion sets for the continuous subcutaneous insulin infusion.
- 1355 If these reactions occur, different adhesives or "under-taping" (such as with IV 3000, Tegaderm,
- etc.) will be tried, sites will be rotated frequently, and a mild topical steroid cream or other
- 1357 medication may be required.
- 1358 Whenever the skin is broken there is the possibility of an infection. The CGM and pump infusion
- sites are inserted under the skin. It is possible that any part that is inserted under the skin may
- cause an infection. These occur very infrequently, but, if an infection was to occur, oral and/or
- topical antibiotics can be used. The risk of skin problems could be greater if you use a sensor for
- longer than it is indicated for use. Therefore, participants will be carefully instructed about proper
- use of the sensor.

#### 1364 **10.2.** Potential Benefits

- 1365 It is expected that this protocol will yield increased knowledge about using a Decision Support
- 1366 System for insulin dosing suggestions. The individual participant may or may not benefit from
- 1367 study participation.

#### 1368 10.3. Risk Assessment

- 1369 Based on the facts that (1) adults with diabetes experience mild hypoglycemia and hyperglycemia
- 1370 frequently as a consequence of the disease and its management, (2) the study intervention
- involves feedback and advice for insulin dosing that may increase the likelihood of hypoglycemia,
- and hyperglycemia, (3) mitigations are in place, and have been tested in prior studies using the
- investigational device system in the home setting. .

#### 1374 **10.4. General Considerations**

- 1375 The study is being conducted in compliance with the policies described in the study policies
- document, with the ethical principles that have their origin in the Declaration of Helsinki, with
- the protocol described herein, and with the standards of Good Clinical Practice (GCP).

DSS-2\_05-Oct-2021 

1378 Whenever possible, data will be directly collected in electronic case report forms, which will be considered the source data.

DSS-2\_05-Oct-2021 

## **Chapter 11 Device Cleaning Instructions**

CGM cleaning instructions are provided in the Dexcom G4 PLATINUM (Professional) Cleaning and Disinfection manual (current edition). The transmitter will be cleaned with Clorox Healthcare® Bleach Germicidal Cleaner or any disinfectant product in a spray bottle containing a bleach solution of 6500 parts per million with the EPA registration number 56392-7. The transmitter will be submerged in this solution and then placed on an absorbent wipe or clean surface. Two sprays will be dispensed from the Clorox cleaner onto each side of the transmitter. A nylon brush will be used to scrub the transmitter on all sides for 30 seconds. The transmitter will be placed in the Clorox Cleaner solution for one minute. The transmitter is then rinsed under flowing tap water for ten seconds. The transmitter will then be disinfected using a disinfectant product with EPA registration number 56392-7 using similar procedures as the cleaning process.

Per the pump manufacturer, the insulin pump will be cleaned with a damp lint-free cloth. Use of household or industrial cleaners, solvents, bleach, scouring pads, chemicals, or sharp instruments are prohibited. The pump should never be submerged in water. If needed, a very mild detergent, such as a bit of liquid soap with warm water will be used. A soft towel will be used to dry the pump.

Equipment that touches intact skin will be cleaned with ethyl or isopropyl alcohol (70-90%), quaternary ammonium germicidal detergent (i.e. Cavicide, EPA number 46781) or household bleach. The contact time on the surface depends on the method used to clean the equipment. Cavicide requires three minutes on the surface of the equipment. Clorox Germicidal Bleach Wipes require two minutes on the equipment. The surface should remain wet (i.e. slightly damp) with the disinfectant to be considered effective though not wet enough to leave drops of liquid.

In the event a manufacturer update for cleaning procedures of their device, the study team will adhere to the most current recommendations.

DSS-2\_05-Oct-2021 

1404

1405

1431

1432

1433

#### 1406 system is experimental. Therefore, an investigational device exemption (IDE) from the U.S. Food and Drug Administration (FDA) is required to conduct the study. 1407 **Definitions** 1408 12.1. 1409 12.1.1. Adverse Events (AE) 1410 A reportable adverse event includes any untoward medical occurrence that meets one of the 1411 following criteria: 1412 A Serious Adverse Event as defined in section 12.1.2 • An Adverse Device Effect as defined in section 12.1.4, unless excluded from reporting in 1413 section 12.8 1414 1415 An Adverse Event as defined in section 12.1.4 occurring in association with a study 1416 procedure • An AE as defined in section 12.1.1 which leads to discontinuation of a study device for 2 1417 1418 or more hours 1419 Hypoglycemia meeting the definition of severe hypoglycemia as defined in section 12.3.1 1420 Diabetic ketoacidosis (DKA) as defined in section 12.3.2 or in the absence of DKA, a 1421 hyperglycemic or ketosis event meeting the criteria defined below 1422 Hypoglycemia and hyperglycemia not meeting the criteria below will not be recorded as adverse 1423 events unless associated with an Adverse Device Effect. Skin reactions from sensor placement 1424 are only reportable if severe and/or required treatment. 1425 12.1.2. Serious Adverse Event (SAE) 1426 Any untoward medical occurrence that: 1427 • Results in death. 1428 Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event). 1429 1430 Requires inpatient hospitalization or prolongation of existing hospitalization.

**Chapter 12 Adverse Events, Device Issues, and Stopping Rules** 

The protocol is considered a significant risk device study due to the fact that the closed loop

DSS-2\_05-Oct-2021 

ability to conduct normal life functions (life threatening).

• Is a congenital anomaly or birth defect.

Results in persistent or significant disability/incapacity or substantial disruption of the

• Is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the participant or may require medical/surgical intervention to prevent one of the outcomes listed above).

#### 1437 12.1.3. Unanticipated Adverse Device Effect (UADE)

- Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of participants (21 CFR 812.3(s)).
- 1443 **12.1.4.** Adverse Device Effect (ADE)
- 1444 Any untoward medical occurrence in a study participant which the device may have caused or to
- which the device may have contributed.
- 1446 **12.1.5. Device Complaints and Malfunctions**
- 1447 A device complication or complaint is something that happens to a device or related to device
- performance, whereas an adverse event happens to a participant. A device complaint may occur
- independently from an AE, or along with an AE. An AE may occur without a device complaint or
- there may be an AE related to a device complaint. A device malfunction is any failure of a device
- 1451 to meet its performance specifications or otherwise perform as intended. Performance
- 1452 specifications include all claims made in the labeling for the device. The intended performance
- of a device refers to the intended use for which the device is labeled or marketed. (21 CFR 803.3).
- 1454 **12.2.** Protocol Deviations
- 1455 A protocol deviation is any noncompliance with the clinical trial protocol, Good Clinical Practices
- 1456 (GCP), or procedure requirements. The noncompliance may be either on the part of the
- participant, the investigator, or the study site staff. As a result of deviations, corrective actions
- 1458 may be developed by the site and implemented as appropriate. Major deviations will be reported
- to the IRB-HSR within 7 calendar days of when the study team becomes aware of the event.
- 1460 **12.3.** Reportable Events
- 1461 **12.3.1.** Hypoglycemia Event
- 1462 Hypoglycemia not associated with an Adverse Device Effect is only reportable as an adverse event
- 1463 when the following definition for severe hypoglycemia is met:

DSS-2\_05-Oct-2021 

1467

1468 1469

1470

1471

1472

1473

1474

1481

1482

1483

1484

1485

1486

1487

1488

1493

- The event required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions;
  - Impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma;
  - If plasma glucose measurements are not available during such an event, neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.

#### 12.3.2. Hyperglycemia Events/Diabetes Ketoacidosis

- Hyperglycemia not associated with an Adverse Device Effect is only reportable as an adverse event when one of the following four criteria is met.
- The event involved DKA, as defined by the Diabetes Control and Complications Trial (DCCT) and described below:
- Evaluation or treatment was obtained at a health care provider facility for an acute event involving hyperglycemia or ketosis
  - Blood ketone level ≥1.5 mmol/L and communication occurred with a health care provider at the time of the event
  - Blood ketone level ≥3.0 mmol/L, even if there was no communication with a health care provider
  - Hyperglycemic events are classified as DKA if the following are present:
    - Symptoms such as polyuria, polydipsia, nausea, or vomiting;
    - Serum ketones ≥1.5 mmol/L or large/moderate urine ketones;
    - Treatment provided in a health care facility
- All reportable Adverse Events—whether volunteered by the participant, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means—will be reported on an adverse event form online. Adverse events will be presented to the DSMB in accumulated manner during each meeting.

#### 12.4. Relationship of Adverse Event to Study Device

1494 The study investigator will assess the relationship of any adverse event to be related or unrelated 1495 by determining if there is a reasonable possibility that the adverse event may have been caused 1496 by the study device.

DSS-2\_05-Oct-2021 

1499

1500

1501

1502

1503

1504

1505

1506 1507

1508

1509

1516

1517

1518

1519

1520

To ensure consistency of adverse event causality assessments, investigators should apply the following general guideline when determining whether an adverse event is related:

- There is a plausible temporal relationship between the onset of the adverse event and the study intervention, and the adverse event cannot be readily explained by the participant's clinical state, intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of response to the study intervention; and/or the adverse event abates or resolves upon discontinuation of the study intervention or dose reduction and, if applicable, reappears upon re-challenge.
- Evidence exists that the adverse event has an etiology other than the study intervention (e.g., preexisting medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the adverse event has no plausible temporal relationship to study intervention.

#### 12.5. Intensity of Adverse Event

- 1510 The intensity of an adverse event will be rated on a three point scale: (1) mild, (2) moderate, or
- 1511 (3) severe. It is emphasized that the term severe is a measure of intensity: thus, a severe adverse
- event is not necessarily serious. For example, itching for several days may be rated as severe, but
- may not be clinically serious.
- MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities.
  - MODERATE: Usually causes a low level of inconvenience or concern to the participant and may interfere with daily activities, but is usually ameliorated by simple therapeutic measures.
  - **SEVERE:** Interrupts a participant's usual daily activities and generally requires systemic drug therapy or other treatment.

#### 1521 **12.6.** Coding of Adverse Events

- 1522 Adverse events will be coded per the UVA IRB website instructions (i.e. mild, moderate, severe).
- 1523 Adverse events that continue after the participant's discontinuation or completion of the study
- 1524 will be followed until their medical outcome is determined or until no further change in the
- 1525 condition is expected.

#### 1526 **12.7.** Outcome of Adverse Events

- 1527 The outcome of each reportable adverse event will be classified by the investigator as follows:
- **RECOVERED/RESOLVED** The participant recovered from the AE/SAE without sequelae.

  Record the AE/SAE stop date.

DSS-2\_05-Oct-2021 

1532

15331534

1535

1536

1537

1538

1539

1540

1541 1542

1543

1544

1545

1546

1547

1548

1549

1550

1551

1552

1553

1554

1555

1561

- **RECOVERED/RESOLVED WITH SEQUELAE** The event persisted and had stabilized without change in the event anticipated. Record the AE/SAE stop date.
  - **FATAL** A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death.
  - **NOT RECOVERED/NOT RESOLVED (ONGOING)** An ongoing AE/SAE is defined as the event was ongoing with an undetermined outcome.
  - An ongoing outcome will require follow-up by the site in order to determine the final outcome of the AE/SAE.
  - The outcome of an ongoing event at the time of death that was not the cause of death, will be updated and recorded as "resolved" with the date of death recorded as the stop date.
  - **UNKNOWN** An unknown outcome is defined as an inability to access the participant or the participant's records to determine the outcome (for example, a participant that was lost to follow-up).

All clinically significant abnormalities of clinical laboratory measurements or adverse events occurring during the study and continuing at study termination should be followed by the participant's physician and evaluated with additional tests (if necessary) until diagnosis of the underlying cause, or resolution. Follow-up information should be recorded on source documents.

If any reported adverse events are present when a participant completes the study, or if a participant is withdrawn from the study due to an adverse event, the participant will be contacted for re-evaluation. If the adverse event has not resolved, additional follow-up will be performed as appropriate. Every effort should be made by the Investigator or delegate to contact the participant until the adverse event has resolved or stabilized.

#### 12.8. Reportable Device Issues

- All UADEs, ADEs, device complaints, and device malfunctions will be reported irrespective of whether an adverse event occurred, except in the following circumstances.
- 1558 The following device issues are anticipated and will not be reported but will reported as an Adverse Event if the criteria for AE reporting described above are met:
- Component disconnections
  - CGM sensors lasting fewer than the number of days expected per CGM labeling
- CGM tape adherence issues

DSS-2\_05-Oct-2021 

1593

1594

Charter.

1563 Pump infusion set occlusion not leading to ketosis 1564 Battery lifespan deficiency due to inadequate charging or extensive wireless 1565 communication 1566 Intermittent device component disconnections/communication failures not leading to 1567 system replacement 1568 Device issues clearly addressed in the user guide manual that do not require additional 1569 troubleshooting • Skin reactions from CGM sensor placement or pump infusion set placement that do not 1570 1571 meet criteria for AE reporting 1572 12.9. Timing of Event Reporting UADEs must be reported within 10 working days to the FDA after the sponsor first 1573 1574 receives notice of the adverse effect. 1575 Other reportable adverse events, device malfunctions (with or without an adverse event) 1576 and device complaints should be reported promptly, but there is no formal required reporting period. 1577 1578 The IDE Sponsor will investigate the UADE and if indicated, report the results of the 1579 investigation to the IRBs, FDA, and DSMB will within 10 working days of the study team becoming aware of the UADE per 21CFR 812.46(b). 1580 1581 • The DSMB will determine if the UADE presents an unreasonable risk to participants. If so, the DSMB will must ensure that all investigations, or parts of investigations presenting 1582 1583 that risk, are terminated as soon as possible but no later than 5 working days after the 1584 DSMB will makes this determination and no later than 15 working days after first receipt notice of the UADE. 1585 1586 • In the case of a device system component malfunction (e.g. pump, CGM, control 1587 algorithm), information will be forwarded to the responsible manufacturer by the study 1588 personnel. 12.10. Data and Safety Monitoring Board 1589 1590 An independent Data and Safety Monitoring Board (DSMB) will be establish to review compiled 1591 safety data at periodic intervals to oversee and monitor our randomized clinical trial to ensure 1592 the safety of participants, as well as the validity and integrity of the data.

DSS-2\_05-Oct-2021 

Details regarding membership, meetings, responsibilities will be documented in a separate DSMB

1617

1618

1619

Medical Monitor document.

#### 1595 12.11. Stopping Criteria 1596 12.11.1. Participant Discontinuation 1597 Rules for discontinuing study device use are: The investigator believes it is unsafe for the participant to continue on the intervention. 1598 1599 This could be due to the development of a new medical condition or worsening of an 1600 existing condition; or participant behavior contrary to the indications for use of the device 1601 that imposes on the participant's safety 1602 The participant requests that the treatment be stopped 1603 Two distinct episodes of DKA 1604 Two distinct severe hypoglycemia events as defined in section 12.3.1 1605 12.11.2. Suspending/Stopping Overall Study 1606 In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or severe 1607 hyperglycemia event, use of the study device system will be suspended while the problem is 1608 diagnosed. 1609 In addition, study activities could be similarly suspended if the manufacturer of any constituent 1610 study device requires stoppage of device use for safety reasons (e.g. product recall). The affected 1611 study activities may resume if the underlying problem can be corrected by a protocol or system modification that will not invalidate the results obtained prior to suspension. 1612 12.12. Independent Safety Oversight 1613 A Medical Monitor will review all DKA and severe hypoglycemia irrespective of relatedness to 1614 study device use, and all serious events (including UADEs) related to study device use at the time 1615 1616 of occurrence. The Medical Monitor can request modifications to the study protocol or

DSS-2\_05-Oct-2021 

suspension or outright stoppage of the study if deemed necessary based on the totality of safety

data available. Details regarding Medical Monitor review will be documented in a separate

1620

# 13.1. Prohibited Medications, Treatments, and Procedures Participants using glulisine at the time of enrollment will be asked to contact their personal physician to change their prescribed personal insulin to lispro or aspart for the duration of the trial. The study devices (study insulin pump, study CGM) must be removed before Magnetic Resonance

- 1626 Imaging (MRI), Computed Tomography (CT) or diathermy treatment. Participants may continue
- in the trial after temporarily discontinuing use if requiring one of the treatments above.

#### 1628 **13.2. Participant Withdrawal**

- Participation in the study is voluntary. Participant may withdraw at any time. For participants who do withdraw from the study, the study team will determine if their data will be used in
- 1631 analysis.

**Chapter 13 Miscellaneous Considerations** 

#### 1632 **13.3. Confidentiality**

For security and confidentiality purposes, subjects will be assigned an identifier that will be used instead of their name. Protected health information gathered for this study may be shared with the third-party collaborators. De-identified subject information may also be provided to collaborators involved in the study after the appropriate research agreement has been executed.

DSS-2\_05-Oct-2021 

1637

1659

1662

## **Chapter 14 Statistical Consideration**

#### 1638 14.1. **Design and Randomization**

- This is a randomized crossover study in T1DM designed to demonstrate the efficacy of 1639
- 1640 personalized feedback (PF) and decision support (DSS) over sensor-augmented pump (SAM)
- therapy and to establish relationships between the level of glucose variability (GV) control 1641
- 1642 achievable by the intervention and individual psycho-behavioral characteristics.
- 1643 We plan to split the study into 4 cohorts of about 25 participants each (expected retention 20
- 1644 per cohort). Each cohort will continue for ~7 months and will have the structure presented in
- 1645 Figure 5. Following recruitment, screening, and a run-in period of SAM, participants will be
- 1646 randomized into one of two groups: escalation vs. de-escalation of devices and function. Each
- 1647 treatment modality (SAM, PF, DSS) will continue for about 8 weeks, with the last 4 weeks used
- to assess GV from CGM data. 1648
- 1649 Escalation: SAM  $\rightarrow$  PF  $\rightarrow$  DSS
- 1650 De-escalation: DSS  $\rightarrow$  PF  $\rightarrow$  SAM
- 1651 14.2. Sample Size

#### 1652 14.2.1. Sample Size Determination:

- 1653 Sample size determination is based on our related pilot studies of DSS. We estimate that the
- 1654 effect size of DSS vs. SAM will be  $f^3$ 0.22. Power calculations (G\*Power 3.1.9.2) assuming a=0.017
- 1655 (corrected for multiple comparisons), 95% power, correlation of 0.55 between the repeated
- measures, and attrition of 20%, yield a sample size of N=100 subjects to be randomized at 1656
- 1657 baseline, with N=80 subjects completing the study. PF vs. SAM assumes the same effect size. We
- expect that while overall DSS effect vs. PF will be smaller than vs. SAM, GV control over time will 1658

be more consistent. Aim 1.3 analysis therefore assumes a small effect size (0.15) but 5 repeated

- 1660 measures (bi-weekly) in each condition with higher correlation (0.65), leading to an achieved
- 1661 power of 97.2% for this Aim.

#### 14.2.2. Exploration of the effect of treatment escalation vs. de-escalation:

- 1663 A key advantage of the proposed study design (beyond the optimal statistical power) is the
- 1664 possibility to explore the glucose control and psycho-behavioral impact of features being added
- 1665 and/or enhanced with prescriptive components (DSS), vs. features being limited to information
- 1666 (PF) or even removed (SAM). We will perform this analysis by looking at the between factors in
- the repeated ANOVA analysis, contrasting the escalation group vs. de-escalation group. While 1667

DSS-2 05-Oct-2021 

- 1668 not powered, this analysis will provide key insights in the future feature adaptation schemes
- 1669 based on the ATI.
- 1670 14.3. **Outcome Measures**
- 1671 14.3.1. Glycemic outcomes:
- The primary outcome of this study will be Glucose Variability (GV) as measured by CGM-based 1672
- 1673 Coefficient of Variation (CV), as recommended by the International Consensus on Use of
- Continuous Glucose Monitoring. To further characterize glucose control, we will compute other 1674
- 1675 CGM Consensus outcomes as well:
- 1676 Average

1679

1680

- Percent in different ranges: 1677
- <50 mg/dL</p> 1678
  - o <54 mg/dL
  - o <60 mg/dL
- o <70 mg/dL 1681
- 1682
- 1683 o >180 mg/dL
- 1684 o >250 mg/dL
- 1685 >300 mg/dL
- SD and coefficient of variation 1686
- 1687 LBGI, HBGI, ADRR
- 1688 Each modality of treatment will be assessed using the last 4 weeks of CGM recordings, as we
- 1689 expect most of the GV benefits of each intervention to be realized within the first 4 weeks of the
- 1690 intervention, and a minimum of 24 days of data is considered optimal for CGM-based CV
- determination. 1691
- 1692 14.3.2. Glucose Variability Reduction Achieved with CGM-based expert systems:
- 1693 General linear models (GLM) (repeated measures ANOVA) will be used to assess the significance of the differences in average response between SAM, PF, and DSS across appropriate CGM-based
- 1694
- 1695 metrics. The particular design of the clinical study allow for Aims 1.1, 1.2, and 1.3 to each be
- 1696 addressed independently in a randomized crossover analysis, as shown in Figure 4. While the
- 1697 randomized order of the interventions (escalation vs de-escalation) allows for an objective
- 1698 assessment of the average efficacy of each of them, we will introduce the order as a fixed factor 1699 to verify if significant study effects can be detected. Finally, we will study the evolution of GV
- 1700 within each modality period: GV and other CGM-based outcomes will be computed bi-weekly
- 1701 (the minimum length of time for precise GV assessment) and entered in a repeated measures

DSS-2\_05-Oct-2021 

- 1702 GLM analysis; within-subject contrast (linear and polynomial) using 5 repeated measures per
- 1703 condition to explore the evolution of the glycemic outcomes in time; Aim 1.3.

#### 1704 **14.4.** Exploration of the effect of treatment escalation vs. de-escalation

- 1705 A key advantage of the proposed study design (beyond the optimal statistical power) is the
- 1706 possibility to explore the glucose control and psycho-behavioral impact of features being added
- and/or enhanced with prescriptive components (DSS), vs. features being limited to information
- 1708 (PF) or even removed (SAM). We will perform this analysis by looking at the between factors in
- the repeated ANOVA analysis, contrasting the escalation group vs. de-escalation group. While
- 1710 not powered, this analysis will provide key insights in the future feature adaptation schemes
- 1711 based on the ATI.

1712

### 14.5. Psychological and Behavioral Questionnaires

- 1713 *Quantitative* data on usability and satisfaction will be analyzed using simple descriptive statistics.
- 1714 In addition, we will analyze scores from the measures in the psychosocial assessment battery to
- determine if changes occur over time and between groups. Using SPSS 26, we will construct
- 1716 predictive models in the general linear modeling (GLM) framework to examine each set of
- 1717 psychological factors (e.g., INSPIRE survey) over time, and their association with glycemic
- 1718 outcomes. Group assignment and Study Phases will be the primary covariate.

#### 1719 **14.6.** Baseline Descriptive Statistics

- 1720 Baseline demographic and clinical characteristics of the cohort of all randomized participants will
- be summarized in a table using summary statistics appropriate to the distribution of each
- variable. Descriptive statistics will be displayed overall and by treatment group.
- 1723 Will include:
- 1724 Age
- HbA1c collected at randomization and study end
- 1726 Gender
- 1727 Race/ethnicity
- CGM use before enrollment
- Diabetes duration
- 1730 BMI

#### 1731 **14.7. Device Issues**

- 1732 We will count each time the participant interacted with the study Personalized Feedback and
- 1733 Decision Support System and perform a Wilcoxon paired rank test to determine if any differences
- 1734 exist in system interactions.

DSS-2\_05-Oct-2021 

# 1735 Chapter 15 Data Collection and Monitoring

#### 1736 **15.1.** Case Report Forms and Device Data

- 1737 The study data are collected through a combination of case report forms (electronic and paper)
- 1738 and electronic device data files obtained from the software and individual hardware
- 1739 components. These electronic device files and electronic CRFs are considered the primary source
- 1740 documentation.
- 1741 When data are directly collected in electronic case report forms, this will be considered the
- source data. Records will be maintained in accordance with ICH E6 and institutional regulatory
- requirements for the protection of confidentiality of participants.

#### 1744 **15.2.** Study Records Retention

- 1745 Study documents will be retained for a minimum of 2 years after study close out. These
- documents may be retained for a longer period, however, if required by local regulations. No
- 1747 records will be destroyed without the consent of the Principal Investigator. It is the responsibility
- of the Principal Investigator to inform all co-investigators when these documents no longer need
- 1749 to be retained.

DSS-2\_05-Oct-2021 

## **Chapter 16 Ethics/Protection of Human Participants**

#### 1751 **16.1. Ethics Standard**

1750

1762

- 1752 The investigator will ensure that this study is conducted in full conformity with Regulations for
- the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21
- 1754 CFR Part 56, and/or the ICH E6.

#### 1755 **16.2.** Institutional Review Boards

- 1756 The protocol, informed consent form(s), recruitment materials, and all participant materials will
- be submitted to the IRB for review and approval. Approval of both the protocol and the consent
- 1758 form must be obtained before any participant is enrolled. Any amendment to the protocol will
- 1759 require review and approval by the IRB before the changes are implemented to the study. All
- 1760 changes to the consent form will be IRB approved; a determination will be made regarding
- whether previously consented participants need to be re-consented.

#### 16.3. Informed Consent Procedures and Documentation

- 1763 Informed consent is a process that is initiated prior to an individual's agreement to participate in
- the study and continues throughout the individual's study participation. Extensive discussion of
- 1765 risks and possible benefits of participation will be provided. Consent forms will be IRB approved
- and the participant will be asked to read and review the document. The investigator or their
- 1767 delegate will explain the research study to the participant and answer any questions that may
- 1768 arise. All participants will receive a verbal explanation in terms suited to their comprehension of
- the purposes, procedures, and potential risks of the study and of their rights as research
- 1770 participants. Participants will have the opportunity to carefully review the written consent form
- 1771 and ask questions prior to signing.
- 1772 The participant will sign the informed consent document prior to any procedures being done
- 1773 specifically for the study. A copy of the informed consent document will be given to the
- participant for their records. The rights and welfare of the participants will be protected by
- emphasizing to them that the quality of their medical care will not be adversely affected if they
- 1776 decline to participate in this study.

#### 1777 16.4. Participant and Data Confidentiality

- 1778 The study monitor, representatives of the IRB or device company supplying study product may
- inspect all documents and records required to be maintained by the investigator, including but
- 1780 not limited to, medical records (office, clinic, or hospital) for the participants in this study.

DSS-2\_05-Oct-2021 

| 1781 | The study participant's contact information will be securely stored at the clinical site for internal |
|---|---|
| 1782 | use during the study. At the end of the study, all records will continue to be kept in a secure |
| 1783 | location for as long a period as dictated by local IRB and Institutional regulations. |
| 1784 | Study participant research data, which is for purposes of statistical analysis and scientific |
| 1785 | reporting, will be stored at the University of Virginia Center for Diabetes Technology. The study |
| 1786 | data entry and study management systems used by research staff will be secured and password |
| 1787 | protected. At the end of the study, all study databases may be de-identified and archived at the |
| 1788 | University of Virginia Center for Diabetes Technology. |

DSS-2\_05-Oct-2021 

## **Chapter 17 References**

- 1790 1. American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes care. 2014 Jan 1;37(Supplement 1): S81-90.
  - 2. Hirsch IB. Insulin analogues. New England Journal of Medicine. 2005 Jan 13;352(2):174-83.
  - 3. Klonoff DC, Prahalad P. Performance of cleared blood glucose monitors. Journal of diabetes science and technology. 2015 Jun 30;9(4):895-910.
  - 4. Castle JR, Jacobs PG. Nonadjunctive use of continuous glucose monitoring for diabetes treatment decisions. Journal of diabetes science and technology. 2016 Sep;10(5):1169-73.
  - 5. Diabetes Control and Complications Trial. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;2005(353):2643-53.
  - 6. Secrest AM, Becker DJ, Kelsey SF, LaPorte RE, Orchard TJ. All-cause mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes. Diabetes care. 2010 Dec 1;33(12):2573-9.
  - 7. Lind M, Svensson AM, Kosiborod M, Gudbjörnsdottir S, Pivodic A, Wedel H, Dahlqvist S, Clements M, Rosengren A. Glycemic control and excess mortality in type 1 diabetes. New England Journal of Medicine. 2014 Nov 20;371(21):1972-82.
  - 8. Nishimura R, LaPorte RE, Dorman JS, Tajima N, Becker D, Orchard TJ. Mortality trends in type 1 diabetes. Diabetes care. 2001 May 1;24(5):823-7.
  - 9. McCall AL, Kovatchev BP. The Median is Not the Only Message: A Clinician's Perspective on Mathematical Analysis of Glycemic Variability and Modeling in Diabetes Mellitus. *J Diabetes Sci Technol* 3: 3-11, 2009.
  - 10. Lachin JM, Genuth S, Nathan DM, Zinman B, Rutledge BN, DCCT/EDIC Research Group: Effect of Glycemic Exposure on the Risk of Microvascular Complications in the Diabetes Control and Complications Trial Revisited. *Diabetes*, <u>57</u>: 995-1001, 2008.
  - 11. Santiago JV. Lessons from the Diabetes Control and Complications Trial, *Diabetes*, 42:1549-1554, 1993.
  - 12. The Diabetes Control and Complications Trial Research Group. The effect of intensive treatment of diabetes on the development and progression of long-term complications of insulin-dependent diabetes mellitus. *N Engl J Med* 329: 978-986, 1993.
  - 13. UK Prospective Diabetes Study Group (UKPDS). Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes. *Lancet* 352: 837-853, 1998.
  - 14. American Diabetes Association Workgroup on Hypoglycemia (Childs BP, Clark NG, Cox DJ, Cryer PE, Davis SN, Di-Nardo MM, Kahn R, Kovatchev BP, Shamoon H). Defining and Reporting Hypoglycemia in Diabetes. *Diabetes Care*, 28:1245-1249, 2005.
- 15. Cryer PE, Davis SN, Shamoon H. Hypoglycemia in Diabetes. *Diabetes Care*, 26: 1902-1912, 2003.

DSS-2\_05-Oct-2021 

- 16. The Diabetes Control and Complications Trial Research Group. Hypoglycemia in the Diabetes Control and Complications Trial. *Diabetes* 46: 271-286, 1997.
- 17. Cryer PE. Hypoglycaemia: The limiting factor in the glycaemic management of type I and type II diabetes. *Diabetologia* 45: 937-948, 2002.
  - 18. Cryer PE: Hypoglycemia: The Limiting factor in the management of IDDM. *Diabetes* 43: 1378-1389, 1994.
  - 19. The Diabetes Control and Complications Trial Research Group: The relationship of glycemic exposure (HbA1c) to the risk of development and progression of retinopathy in the Diabetes Control and Complications Trial. *Diabetes* 44:968–983, 1995.
  - 20. Brownlee M, Hirsh IB. Glycemic Variability: A hemoglobin A1c–Independent Risk Factor for Diabetic Complication? *JAMA*, <u>295</u>: 1707-1708, 2006.
  - 21. Hirsh IB, Brownlee M: Should minimal blood glucose variability become the gold standard of glycemic control? *J Diabetes Complications*, <u>19</u>:178–181, 2005.
  - 22. Esposito K, Giugliano D, Nappo F, Martella K, for the Campanian Postprandial Hyperglycemia Study Group. Postprandial Hyperglycemia Study Group. Regression of carotid atherosclerosis by control of postprandial hyperglycemiain type 2 diabetes mellitus. *Circulation* 110: 214-219, 2004.
  - 23. Haffner S.M. The importance of postprandial hyperglycaemia in development of cardiovascular disease in people with diabetes: *International Journal of Clinical Practice*. Supplement 123: 24-26, 2001.
  - 24. Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of Oxidative Stress by Acute Glucose Fluctuations Compared With Sustained Chronic Hyperglycemia in Patients With Type 2 Diabetes. *JAMA* 2006 295: 1681-1687.
  - 25. Temelkova-Kurktschiev TS, Koehler C, Henkel E, Leonhardt W, Fuecker K, Hanefeld M. Postchallenge Plasma Glucose and Glycemic Spikes are More Strongly Associated With Atherosclerosis Than Fasting Glucose or HbA1c Level. *Diabetes Care*, 23:1830–1834, 2000.
  - 26. Waldhäusl WK. The physiological basis of insulin treatment—clinical aspects. Diabetologia. 1986 Dec 1;29(12):837-49.
  - 27. Grunberger G, Abelseth JM, Bailey TS, et al Consensus statement by the American Association of Clinical Endocrinologists/American College of Endocrinology Insulin Pump Management Task Force. Endocr Pract 2014;20:463–89.
  - 28. YB Kim and J. Lee, "Smart Devices for Older Adults Managing Chronic Disease: A Scoping Review," JMIR Mhealth and Uhealth, 5(5):e69, 2017.
  - 29. K. Singh, K. Drouin, L. P. Newmark, et al., "Patient-Facing Mobile Apps to Treat High-Need, High-Cost Populations: A Scoping Review," JMIR Mhealth and Uhealth, 4(4):e316, 2016.
  - 30. N. Kaufman and A. Salahi, "Using Digital Health Technology to Prevent and Treat Diabetes," Diabetes Technology & Therapeutics, 19(Supplement 1):59-73.
  - 31. H. D. Lehmkuhl et al., "Telehealth Behavior Therapy for the Management of Type 1 Diabetes in Adolescents," J. Diabetes Science and Technology, 4(1):199-208, 2010.

DSS-2\_05-Oct-2021 

- 32. C. L. Wood, et al., "Use of Telemedicine to Improve Adherence to American Diabetes
   Association Standards in Pediatric Type 1 Diabetes," Diabetes Technology & Therapeutics,
   18(1):7-14, 2016.
- 1871 33. B. P. Kovatchev, P. Mendosa, S. Anderson, J. S. Hawley, L. M. Ritterband, L. Gonder-1872 Frederick, "Effect of Automated Bio-Behavioral Feedback on the Control of Type 1 1873 Diabetes," Diabetes Care, 34:302-307, 2011.
  - 34. D. C. Klonoff and D. Kerr, "Digital Diabetes Communication: There's an App for That," J. Diabetes Science and Technology, 10(5):1003-1005, 2016.
    - 35. H. Zisser, L. Jovanovic, F. J. Doyle III, P. Ospina, and C. Owens. Run-to-run control of meal-related insulin dosing. Diab Technol Ther, 7:48–57, 2005.
    - 36. C. Owens, H. Zisser, L. Jovanovic, B. Srinivasan, D. Bonvin, and F. J. Doyle III. Run-to-run control of blood glucose concentrations for people with type 1 diabetes mellitus. IEEE Trans Biomed Eng, 53:996–1005, 2006
    - 37. P. Herrero, P. Pesl, M. Reddy, N. Oliver, P. Georgiou, and C. Toumazou. Advanced insulin bolus advisor based on run-to-run control and case-based reasoning. IEEE Journal of Biomedical and Health Informatics, 19(3):1087–1096, 2015.
    - 38. C.C. Palerm, H. Zisser, W.C. Bevier, L. Jovanovic, and F. J. Doyle III. Prandial insulin dosing using run-to-run control: application of clinical data and medical expertise to define a suitable performance metric. Diabetes Care, 30:1131–1136, 2007.
    - 39. C.C. Palerm, H. Zisser, L. Jovanovic, and F. J. Doyle III. A run-to-run control strategy to adjust basal insulin infusion rates in type 1 diabetes. J Process Control, 18:258–265, 2008.
    - 40. L. Kennedy and A. Brown, "FDA Clears 'My Dose Coach' App to Optimize Basal Insulin Dosing," diaTribe: Making Sense of Diabetes, (https://diatribe.org/fda-clears-my-dose-coach-app-to-optimize-basal-insulin-dosing), posted April 2017.
    - 41. S. D. Patek, D. Lv, E. Campos-Nanez, M. Breton, "Retrospective Optimization of Daily Insulin Therapy Parameters: Control Subject to a Regenerative Disturbance Process," IFAC Symposium on Dynamics and Control of Process Systems, IFAC-PapersOnLine 49-7, pp. 773-778, 2016.
    - 42. C. Toffanin, A. Sandri, M. Messori, C. Cobelli, and L. Magni. Automatic adaptation of basal therapy for type 1 diabetic patients: a run-to-run approach. In IFAC 19th World Congress, pages 2070–2075, 2014.
    - 43. Steil GM, Oladunjoye AO, Wald JS, Slyne C, Atakov-Castillo A, Greenberg J, Greaves T, Toschi E, Munshi M. Use of Automated Clinical Decision Support (CDS) to Effect Glycemic Control in Elderly Patients with T1D.
    - 44. J. Tuo et al., "Optimization of insulin pump therapy based on high order run-to-run control scheme," Comput Methods Programs Biomed, 120(123-134), 2015.
    - 45. Doyle FJ, 3rd, Huyett LM, Lee JB, Zisser HC, Dassau E. Closed-loop artificial pancreas systems: engineering the algorithms. Diabetes care 2014;37:1191-7.
  - 46. Hovorka, R et al. Manual closed-loop insulin delivery in children and adolescents with Type 1 Diabetes: A phase 2 randomised crossover trial. *The Lancet*, **375**, 743-751 (2010).

DSS-2\_05-Oct-2021 

- 47. Anderson SM et al. Multinational Home Use of Closed-Loop Control Is Safe and Effective.
   Diabetes Care 39, 1143-1150 (2016).
  - 48. B.P. Kovatchev, E. Renard, C. Cobelli, et al. "Feasibility of outpatient fully integrated closed-loop control: first studies of wearable artificial pancreas", Diabetes Care, 36(7):1851-8, 2013
  - 49. P. Keith-Hynes, B. Mize, A. Robert and J. Place, "The diabetes assistant: a smartphone-based system for real-time control of blood glucose", Electronics, 3(4):609-623, 2014
  - 50. J. Place, A. Robert, N.B. Brahim, et al. "DiAs web monitoring: A real-time remote monitoring system designed for artificial pancreas outpatient trials", J. Diabetes Sci. Technol., 7(6):1427-1435, 2013
  - 51. Lau, N, McElwee M, Wakeman C, DeBoer M, Chernavvsky DR, Real Time Remote Monitoring with Artificial Panrceas: A Family-Centered Pilot Trial, Diabetes Care 63 Sup 1: LB27, 2014
  - 52. Gonder-Frederick L, Hughes-Karvetski C, McElwee M, Kovatchev BP, Interactive Internet Intervention Providing Individually-Tailored Glycemic Feedback Based on CGM, Insulin and Meal Data, and Computer Simulation: Content Design. Diabetes Technology & Therapeutics. February 2013, 15(S1): A-104-A-105
  - 53. Kubiak T, Mann CG, Barnard KD and Heinemann L. Psychosocial Aspects of Continuous Glucose Monitoring: Connecting to the Patients' Experience. J Diabetes Sci Technol 2016 Jul; 10(4): 859-863
  - 54. Barnard KD and Weisberg-Benchell J, Psychosocial Aspects and Diabetes Technology: Head to Head or Hand in Hand. European Endocrinology 12(1):35 January 2016
  - 55. Friedman B, Kahn PH, Howe JR and Howe DC 2000. Trust online, Communications of the ACM, 43, 12, 34-40.
  - 56. Ritholz MD, Atakov-Castillo A, Beste M, et al. Psychosocial factors associated with use of continuous glucose monitoring. Diabet Med. 2010;27:1060-1065
  - 57. Lieberman A, Barnard K. Diabetes technology and the human factor. Diabetes Technology & Therapeutics. Feb 2018.S-128-S-138.http://doi.org/10.1089/dia.2018.2511
  - 58. Barnard KD, Wysocki T, Thabit H, Evans M et al. Psychosocial Aspects of Closed and Open Loop Insulin Delivery: Closing the Loop In Adults with Type 1 Diabetes in the Home Setting Diabetic Medicine 32(5) January 2015 DOI: 10.1111/dme.12706
  - 59. Kovatchev BP, Patek SD, Dassau E, Doyle FJ III, Magni L, De Nicolao G, and Cobelli C. Control-to-range for diabetes: functionality and modular architecture, J Diabetes Sci Technol, 3: 1058-1065, 2009.
  - 60. Patek SD, Magni L, Dassau E, Karvetski CH, Toffanin C, DeNicolao G, DelFaverokS, Breton M, Dalla Man C, Renard E, Zisser H, Doyle FJ III, Cobelli C, Kovatchev BP. Modular Closed-Loop Control of Diabetes, Transactions on Biomedical Engineering, 29: 2986-3000, 2012.
  - 61. Kovatchev BP, Cox DJ, Gonder-Frederick LA Young-Hyman D, Schlundt D, Clarke WL. Assessment of risk for severe hypoglycemia among adults with IDDM: Validation of the Low Blood Glucose Index, *Diabetes Care* 21: 1870-1875, 1998.

DSS-2\_05-Oct-2021 

- 1948 62. Brown SA, Jiang B, McElwee-Malloy M, Wakeman C, Breton MD. Fluctuations of 1949 hyperglycemia and insulin sensitivity are linked to menstrual cycle phases in women with 1950 T1DM. Journal of diabetes science and technology. 2015 Oct 14;9(6):1192-9.
  - 63. Swan KL, Dziura JD, Steil GM, Voskanyan GR, Sikes KA, Steffen AT, Martin ML, Tamborlane WV, Weinzimer SA. Effect of age of infusion site and type of rapid-acting analog on pharmacodynamic parameters of insulin boluses in youth with type 1 diabetes receiving insulin pump therapy. Diabetes Care. 2009 Feb 1;32(2):240-4.
  - 64. Ben Brahim N, Place J, Renard E, Breton MD. Identification of main factors explaining glucose dynamics during and immediately after moderate exercise in patients with type 1 diabetes. Journal of diabetes science and technology. 2015 Oct 18;9(6):1185-91.
  - 65. Kovatchev BP. Metrics for glycaemic control from HbA1c to continuous glucose monitoring. Nature Reviews Endocrinology. 2017 Jul 1;13(7):425-36.
  - 66. Cox, DJ, Carter, WR, Gonder-Frederick, LA, Clarke, WL, Pohl, S. Blood Glucose Discrimination Training in Insulin-Dependent Diabetes Mellitus Patients. Biofeedback and Self-Regulation. 1988;13(3):201-217.
  - 67. Cox, DJ, Gonder-Frederick, LA, Julian, D, Cryer, P, Lee, JH, Richards, FE, Clarke, WL. Intensive Versus Standard Blood Glucose Awareness Training (BGAT) with Insulin-Dependent Diabetes: Mechanisms and Ancillary Effects. Psychosomatic Medicine. 1991;53(4):453-462.
  - 68. Cox, DJ, Gonder-Frederick, LA, Julian, D, Clarke, W. Long-term Follow-up Evaluation of Blood Glucose Awareness Training. Diabetes Care. 1994;17(1):1-5.
  - 69. Cox, D, Gonder-Frederick, L, Polonsky, W, Schlundt, D, Julian, D, Clarke, W. A Multicenter Evaluation of Blood Glucose Awareness Training-II. Diabetes Care. 1995;18(4):523-8.
  - 70. Gonder-Frederick LA, Julian DM, Cox DJ, Clarke WL, Carter WR. Self-measurement of blood glucose: Accuracy of self-reported data and adherence to recommended regimen. Diabetes Care. 1988;11(7):579-585.
  - 71. Gonder-Frederick LA, Cox DJ, Bobbitt SA, Pennebaker JW. Mood changes associated with blood glucose fluctuations in insulin dependent diabetes mellitus. Health Psychology. 1989;8(1):45-59.
  - 72. Clarke WL, Cox DJ, Gonder-Frederick LA, Julian D, Schlundt D, Polonsky W. The relationship between non-routine use of insulin, food and exercise and the occurrence of hypoglycemia in adults with IDDM and varying degrees of hypoglycemic awareness and metabolic control. Diabetes Educator. 1997;23(1):55-58.
  - 73. Clarke WL, Cox DJ, Gonder-Frederick LA, Julian D, Kovatchev B, Young-Hyman D. The biopsychobehavioral model of risk of severe hypoglycemia II: Self-management behaviors. Diabetes Care. 1999;22(4):580-584.
  - 74. Clarke WL, Cox DJ, Gonder-Frederick LA, Kovatchev B. Hypoglycemia and the decision to drive a motor vehicle by persons with diabetes. JAMA. 1999;282(8):750-4.
  - 75. Cox DJ, Gonder-Frederick LA, Schroeder DB, Cryer PE, Clarke WL. Disruptive effects of acute hypoglycemia on speed of cognitive and motor performance. Diabetes Care. 1993;16(10):1391-1393.

DSS-2\_05-Oct-2021 

- 76. Cox DJ, Kovatchev BP, Gonder-Frederick LA, Summers K, McCall A, Grimm KJ, Clarke WL.
  Relationships between hyperglycemia and cognitive performance among adults with type
  1 and type 2 diabetes mellitus. Diabetes Care. 2005;28(1):71-77.
  - 77. Cox D, Gonder-Frederick L, McCall A, Kovatchev B, Clarke W. The effects of glucose fluctuation on cognitive function and QOL: the functional costs of hypoglycaemia and hyperglycaemia among adults with type 1 or type 2 diabetes. International journal of clinical practice. Supplement. 2002;(129):20-6.
  - 78. Gonder-Frederick L, Zrebiec J, Bauchowitz A, Lee J, Cox D, Ritterband L, Kovatchev B, Clarke W. Detection of hypoglycemia by children with type 1 diabetes 6 to 11 years of age and their parents: a field study. Pediatrics. 2008;121(3):e489-95.
  - 79. Gonder-Frederick, LA, Zrebiec, JF, Bauchowitz, AU, Ritterband, L, Magee, JC, Cox, DJ, Clarke WL. Cognitive Function Is Disrupted by Both Hypo-and Hyperglycemia in School-Aged Children With Type 1 Diabetes: A Field Study. Diabetes care. 2009;32(6):1001-6.
  - 80. Gonder-Frederick LA, Grabman JH, Kovatchev, B, Brown SA, Patek S, Basu A, Pinsker JE, Kudva YC, Wakeman CA, Dassau E, Cobelli C. Is Psychological Stress a Factor for Incorporation into Future Closed-Loop Systems? Journal of Diabetes Science and Technology. 2016;10(3)640-6.
  - 81. Gonder-Frederick LA, Grabman JH, Shepard JA, Tripathi AV, Ducar DM, McElgunn ZR. Variability of Diabetes Alert Dog Accuracy in a Real-World Setting. Journal of Diabetes Science and Technology. 2017;doi: 1932296816685580.
  - 82. Gonder-Frederick LA, Grabman, JH, Shepard JS. Diabetes Alert Dogs (DADs): An Assessment of Accuracy and Implications. Diabetes Research and Clinical Practice Volume 134, December 2017, Pages 121-130
  - 83. Jackson DN, & Tremblay PF. The Six-Factor Personality Questionnaire. In B. de Raad & M. Perugini (Eds.), Big Five Assessment (p. 354-372). Hogrefe & Huber Publishers.
  - 84. Ziegler R, Cavan DA, Cranston I, Barnard K, Ryder J, Vogel C, Parkin CG, Koehler Vesper I, Petersen B, Schweitzer MA, Wagner RS. Use of an Insulin Bolus Advisor Improves Glycemic Control in Multiple Daily Insulin Injection (MDI) Therapy Patients With Suboptimal Glycemic Control. Diabetes Care. 2013 Nov 36(11) 3613-3619.
  - 85. Peyrot M, Rubin RR. Structure and Correlates of Diabetes-Specific Locus of Control. Diabetes Care. 1994;17:994–1001.
  - 86. Ferraro LA, Price JH, Desmond SM, Roberts S. Development of a Diabetes Locus of Control Scale. Psychological Reports, 1987, Volume: 61 (3) 763-770.
  - 87. Van Der Ven NC, Weinger K, Yi J, Pouwer F, Adèr H, Van Der Ploeg HM, Snoek FJ. The Confidence in Diabetes Self-Care Scale: Psychometric Properties of a New Measure of Diabetes-Specific Self-Efficacy in Dutch and US Patients with Type 1 Diabetes. Diabetes Care. 2003;26(3):713–718. doi:10.2337/diacare.26.3.713
  - 88. Clarke WL, Cox DJ, Gonder-Frederick LA, Julian D, Schlundt D, Polonsky W. Reduced Awareness of Hypoglycemia in Adults with IDDM: A Prospective Study of Hypoglycemic Frequency and Associated Symptoms. Diabetes Care 18:517–522, 1995

DSS-2\_05-Oct-2021 

2032

20332034

2035

2036

2037

2038

20392040

2041

20422043

2044

20452046

20472048

2049

- 89. Fisher L, Hessler DM, Polonsky WH, Mullan J. (2012). When is Diabetes Distress Clinically Meaningful? Establishing Cut-Points for the Diabetes Distress Scale. Diabetes Care, 35, 259-264.
  - 90. Polonsky WH, Fisher L, Esarles J, Dudl RJ, Lees J, Mullan JT, Jackson R (2005). Assessing Psychosocial Distress in Diabetes: Development of the Diabetes Distress Scale. Diabetes Care, 28, 626-631.
  - 91. Gonder-FrederickLA, Schmidt KM, Vajda KA, et al. Psychometric Properties of the Hypoglycemia Fear Survey-ii for Adults with Type 1 Diabetes. Diabetes Care. 2011;34(4):801–806, 2011.
  - 92. Singh H, Gonder-Frederick L, Schmidt K, Ford D, Vajda KA, Hawley, Cox DJ. Assessing Hyperglycemia Avoidance in People with Type 1 Diabetes. Diabetes Management. 4(3):263-271, 2014.
  - 93. Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: A New Instrument for Psychiatric Practice and Research. Psychiatry Res. 1988;28:193–213. PMID: 2748771 DOI:10.1016/0165-1781(89)90047-4
  - 94. Weissberg-Benchell J, Hessler D, Polonsky WH, Fisher L. Psychosocial Impact of the Bionic Pancreas During Summer Camp. J Diabetes Sci Technol. 2016;10(4):840–844, 2016.
  - 95. Weissberg-Benchell J, Shapiro JB, Hood K, Laffel LM, Naranjo D, Miller K, Barnard K. Assessing patient-reported outcomes for automated insulin delivery systems: the psychometric properties of the INSPIRE measures. Diabet Med. 2019 May;36(5):644-652. doi: 10.1111/dme.13930.

DSS-2\_05-Oct-2021 